Official Title:

Local Open-label Multicenter Study to Assess the Effectiveness of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis in Russian

Clinical Practice

NCT03208933 NCT Number:

**Document Date:** SAP Version 2.0: 17-Jun-2020

# Data MATRIX

SF\_STAT001\_ver 2\_Eag Approval Date 19 July 2017

## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.8\_17 June 2028

Protocol Number: ML39355

Protocol Title:

LOCAL OPEN-LABEL MULTICENTER STUDY TO ASSESS THE EFFECTIVENESS OF PIRFENIDONE IN PATIENTS WITH IDIOPATHIC PULMONARY FIBROSIS IN RUSSIAN CLINICAL

PRACTICE

SAP version: Final 2.0

Effective date:

17.06.2020





## **Revision History**

| № | Date | Changes Implemented | Version Number |
|---|---|---|---|
| 1 | 22.01.2020 | New document | 1.0 |
| 2 | 17.06.2020 | Section 9.2 (Adverse Events) was updated to include additional adverse event summaries. New tables (3.12.X, 3.13.X, 3.14) were added as requested by Roche Regulatory Disclosures and described in ML39355 Study Results Posting Requirements. The numeration of subsequent tables was adjusted. Section 7 (Summary of Study Data) was updated with the statement regarding summary of data from patients who received different Pirfenidone drugs during rollover study. Numeration of sections was adjusted according to the latest template version. Typing errors were corrected. | 2.0 |



## **Table of Contents**

| | Abbreviations and Definitions | | |
|----|--------------------------------------------------|--------------|---|
| | Introduction | | |
| 3. | Study Objectives and Endpoints | 5 | 5 |
| | 3.1. Study Objectives | 5 | 5 |
| | 3.2. Endpoints | 5 | ; |
| 4. | Study Design | <del>(</del> | 5 |
| | 4.1. General Study Design and Plan | <del>(</del> | 5 |
| | 4.2. Randomization and Blinding | . 11 | ĺ |
| 5. | Sample Size | . 11 | ĺ |
| 6. | General Considerations | . 11 | l |
| | 6.1. Timing of Analyses | . 11 | l |
| | 6.2. Analysis Populations | . 12 | 2 |
| | 6.3. Missing Data | . 12 | 2 |
| | 6.4. Interim Analyses and Data Monitoring | . 14 | ļ |
| | 6.5. Multi-center Studies | | |
| | 6.6. Multiple Testing | . 14 | ļ |
| 7. | Summary of Study Data | . 14 | ļ |
| | 7.1. Subject Disposition | | |
| | 7.2. Protocol Deviations | . 16 | 5 |
| | 7.3. Demographic and Baseline Variables | . 17 | 7 |
| | 7.4. Concurrent Illnesses and Medical Conditions | | |
| | 7.5. Prior and Concurrent Medications | | |
| 8. | Efficacy Analyses | | |
| | 8.1. Primary Efficacy Analysis | | |
| | 8.2. Secondary Efficacy Analyses | | |
| | 8.3. Exploratory Efficacy Analyses | | |
| 9. | Safety Analyses | | |
| | 9.1. Exposure | | |
| | 9.2. Adverse Events | | |
| | 9.3. Pregnancies | | |
| | 9.4. Clinical Laboratory Evaluations | | |
| | 9.5. Other Safety Measures | | |
| 1( | ). Pharmacokinetics | | |
| | Other Analyses | | |
| | . Reporting Conventions | | |
| | Technical Details | | |
| | Summary of Changes to the Protocol | | |
| | . References | | |
| 16 | 5. Listing of Tables, Listings and Figures | . 30 | ) |
| | 16.1. Tables | | |
| | Patients Disposition | | |
| | Protocol Deviations | | |
| | Demographic and Anthropometric characteristics | | |
| | Baseline Variables | | |
| | Medical history | | |
| | Prior and concomitant medications. | | |
| | Efficacy Analyses | | |
| | Primary Efficacy Endpoint | | |
| | Secondary Efficacy Endpoint | | |
| | Exploratory Efficacy Endpoint | | |
| | Safety Analyses | | |
| | 16.2. Figures | | |
| | 16.3. Listings | | |

## 1. Abbreviations and Definitions

The abbreviations and the definitions used in this document are listed below.

| | definitions used in this document are listed below. |
|---|---|
| Abbreviation | Definition |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| AP | Alkaline phosphatase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Classification |
| ATS | American Thoracic Society |
| BAL | Bronchoalveolar lavage |
| BMI | Body mass index |
| ccs | Complete case set |
| CS | Clinically significant |
| CI | Confidence interval |
| CK | Creatine kinase |
| CSR | Clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLco | Carbon monoxide diffusing capacity |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| CRF | Case Report Form |
| EQ-5D-5 | European Quality of Life 5-Dimension Questionnaire |
| | cluding five levels of severity in each of the existing five EQ- |
| ` | dimensions) |
| FAS | Full analysis set |
| FEV | Forced expiratory volume |
| (F)VC | (Forced) Vital capacity of the lungs |
| FU | Follow up |
| GAP | Gender, Age, Physiology (multidimensional index and |
| | staging system for IPF) |
| GGT | Gamma-glutamyl transferase |
| Hb | Hemoglobin |
| (HR)CT | (High-resolution) Computer Tomography |
| lìch' | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IMP | Investigational Medicinal Product |
| ILD | Interstitial lung disease |
| IPF | Idiopathic Pulmonary Fibrosis |
| LDH | Lactic dehydrogenase |
| LOCF | Last observation carried forward |
| MDT | Multidisciplinary team |
| (n)MWT | N-minute wa k test |
| NCS | Not clinically significant |
| PFT | Pulmonary function test |
| PRO | Patient-reported outcome |
| PT | Preferred term |
| QTC-F | QT interval corrected (using Fridericia's formula) |
| RBC | Red blood cells |
| SAE | Serious Adverse Event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SOC | System organ class |
| SOP | Standard operating procedure |
| SSD | Sum of squared deviations |
| SLB | Surgical lung biopsy |
| TEAE | Treatment emergent adverse events |
| TID | Three times per day |
| TS | Treated set |
| UIP | Usual interstitial pneumonia |
| I - | |



| VAS | Visual Analogue Scale |
|-----|-----------------------|
| WBC | White blood cells |
| yr | Year |

#### 2. Introduction

This SAP is written according to ICH E9 Guideline [1] and Data MATRIX LLC SOP [2, 3] using the Protocol Final version 2.0 dated 01.02.2019 and CRF Final version 1.2 dated 08.07.2019.

The purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis, described in the Protocol, and to include detailed procedures for executing the statistical analysis.

The SAP needs to be finalized and signed prior to database soft lock. Revisions to the approved SAP may be made prior to database soft lock. In case of deviation from the finalized SAP, explanation will be provided in the clinical study report (CSR).

#### 3. Study Objectives and Endpoints

#### 3.1. Study Objectives

## 3.1.1. Primary Efficacy Objective

To estimate the treatment effect of pirfenidone 2403 mg/d on lung function.

#### 3.1.2. Secondary Efficacy Objective

To estimate the effectiveness of pirfenidone on IPF patients' functional capability and quality of life.

#### 3.1.3. Exploratory Efficacy Objective

To estimate the effectiveness of pirfenidone on the frequency and number of acute exacerbations of IPF and on features of HRCT.

#### 3.1.4. Safety Objective

To evaluate the safety of pirfenidone.

#### 3.2. Endpoints

#### 3.2.1. Primary Efficacy Endpoint

 Change from Baseline to Week 26 in absolute mL forced vital capacity (FVC) and % FVC

#### 3.2.2. Secondary Efficacy Endpoints

- Change from baseline to Week 26 in 6-minute walk test (6MWT) distance
- Change from baseline to Week 26 in patients' quality of life as measured with European Quality of Life 5-Dimension Questionnaire (EQ-5D)

#### 3.2.3. Exploratory Efficacy Endpoints

• Frequency and number of IPF exacerbations



• CT scan evaluation (semiquantitative assessment "HRCT fibrosis score". The highresolution computed tomography (HRCT) findings will be evaluated using HRCT scoring system. Interstitial lung disease (ILD) radiologist will make assessment of 4 main findings in three zones of each lung. The six zone scores will be averaged to determine the total score for each patient at baseline and at Weeks 26 and 52)

## 3.2.4. Safety Endpoints

- Treatment-emergent adverse events (AEs)
- Treatment-emergent serious adverse events (SAEs)
- Change from baseline in clinical laboratory parameters and electrocardiogram (ECG) parameters

## 4. Study Design

## 4.1. General Study Design and Plan<sup>1</sup>

This is a local, multicenter, interventional, non-randomized, non-controlled, non-comparative, open-label study to assess the effectiveness of pirfenidone in patients with IPF in Russian clinical practice. Approximately 60 patients diagnosed IPF will be enrolled to receive pirfenidone 2403 mg/d for 26 weeks. No comparator group is implied in the study.

For enrolment into the study, the diagnosis of IPF must be confirmed by central review of HRCT scans and of the surgical lung biopsy (SLB) samples, if available (if performed prior enrolment in routine clinical practice). The HRCT scans will be reviewed by one or two central readers who are radiologists with expertise in IPF. If the first expert (central reader-1) agrees with the local opinion, the second expert (central reader-2) will not review scans. If the first expert disagrees with the local opinion, the second expert should review scans. Histopathological (SLB) samples will be reviewed by the one central reader who is a pathologist with expertise in IPF. All other diagnostic procedures will be performed and assessed at a local level.

Eligible patients aged 40–80 years must have a confident clinical and radiographic/ or histological diagnosis of IPF according to 2011 IPF guidelines (ATS 2011). Patients with possible UIP on high-resolution computed tomography and without SLB in case of "working diagnose" of IPF during multidisciplinary team (MDT) discussion, are also eligible for the trial (see Table 2).

Patients will be required to have a relative %FVC  $\geq$  40 %, percent predicted carbon monoxide diffusing capacity (%DLCO)  $\geq$  30 %, and able to walk  $\geq$  100 meters during the 6-minute walk test at the Screening.

All assessments in the study will be initiated only after signed Informed Consent is obtained from the patient. For this purpose, an additional visit may be performed prior to the start of the Screening procedures and an appropriate review of the patient's clinical data relevant to the IPF diagnosis is done.

Any patient identified for the study must discontinue all prohibited therapies including therapy targeted to treat IPF for at least 28 days before the start of the treatment period. Other than

<sup>&</sup>lt;sup>1</sup> This section is based on the sections 3.1 "Description of the study", 3.2 "End of study and length of study" of the clinical study Protocol.



permanent use of corticosteroids (prednisolone at a maximum daily dose of 15 mg or equivalents) and brief periods of corticosteroid use for acute IPF exacerbation, patients will not receive any other therapy for the treatment of IPF. After central review of HRCT and SLB, patients will enter the Screening period, which may last up to 28 days (4 weeks).

After the Screening, eligible patients will enter the Treatment period lasting  $26 (\pm 1)$  weeks. All patients will receive pirfenidone 2403 mg/d administered orally in divided doses three times per day (TID) with food. Dose of the study treatment will be titrated over 14 days to the full dose of 9 capsules per day (three 267 mg capsules taken orally TID with food). Patients will remain on a stable maintenance dose for the duration of the treatment period unless the dose is reduced to manage adverse events or titrated again when restarting study treatment after an appropriate interruption in treatment.

The primary efficacy endpoint in the study is the change from baseline to Week 26 in absolute (mL) FVC and relative (%) FVC as measured by spirometry procedure. Spirometry will be performed at the Screening, on Day 1 of treatment, at Week 12, Week 26 and in the extended Follow-up period (Weeks 39 and 52), if applicable. At screening, spirometry measurements will be performed before and after administration of albuterol (or salbutamol) from a metered dose inhaler. During further visits, bronchodilator test is not necessary to perform. Spirometry data collected throughout the study will be evaluated by local readers.

Patients will have a telephone assessment at Week 1, when safety-related information and adherence to treatment is collected. Subsequently patients will have in-clinic visits at Weeks 2, 4, 8, 12, 16, 20 and 26. Patients should complete an adverse event and dosing compliance diary between all visits. Additionally, telephone calls to patients will be scheduled at Weeks 3, 5, 7, 13 and 24 as a part of IPF care program. A total of 5-7 calls are scheduled in the study, including extra-calls at Weeks 8 and 10 as needed.

Treatment with pirfenidone will continue until Week  $26 (\pm 1)$ . Patients will be followed through the Follow-up visit scheduled 2-4 weeks after treatment completion or until entry into the long-term follow-up (rollover study), whichever occurs earlier. Patients who undergo lung transplantation or who chose to withdraw from study procedures early will be followed for vital status until Week 26. If patients discontinue study treatment early for any reason, they should continue with all scheduled study procedures through Week 26.

Patients who complete participation in the study prematurely due to any reasons (drop-outs) will not be replaced.

Patients who proceed until Week 26 in the study and are compliant with the study treatment, may continue treatment with commercially available pirfenidone after study completion in real clinical practice (long-term follow-up or rollover study). In this case, patients will have two follow-up assessments of FVC and 6MWT at Weeks 39 and 52 and CT scans evaluation at Week 52. Information on AEs occurrence will also be collected during the rollover part of the study.

If a patient cannot participate in the rollover part of the study for any reason, a follow-up visit will be performed 14-28 days after the last dose of pirfenidone is taken.

A schedule of activities is provided in Table 1.

An Independent Data Monitoring Committee (IDMC) will be implemented in the study. The



IDMC will conduct regular review of the trial safety data, with the focus on death cases, serious adverse events, unexpected adverse events, adverse events leading to treatment or study discontinuation, liver enzyme increases, reported as adverse events, and other AEs immediately reported to the Sponsor.

Duration of participation in the study for an individual patient is between 31 and 35 weeks (excluding long-term follow-up). For patients continuing in the rollover study the duration of participation in the study extends up to maximum 58 weeks.

Table 1 Schedule of Activities

| Study period | IC<br>visit | Screening<br>(Washout, if<br>applicable) | | Treatment period | | | | | | Follow-Up | | -Term<br>w-Up <sup>16</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week/ Day<br>(Window) | | –4 to −1 W | Day 1 | W1<br>(± 1 d) | W2<br>(± 2 d) | W4<br>(± 2 d) | W8<br>(± 2 d) | W12<br>(± 2 d) | W16<br>(± 1 w) | W20<br>(± 1 w) | | 26<br>I w) | 14–28 days<br>after last<br>dose | W39<br>(± 2 w) | W52<br>(± 2 w) |
| Informed consent <sup>1</sup> | X | | | | | | | | | | | | | | |
| Phone Call Assessment <sup>2</sup> | | | | х | | | | | | | | | | | |
| Demographic data | | X | | | | | | | | | | | | | |
| Medical history, concomitant medication <sup>3</sup> | X <sup>3</sup> | X <sup>3</sup> | X | | X | X | x | X | X | X | | X | x | | |
| Vital signs, physical exam <sup>4</sup> | | х | X | | X | х | х | X | X | X | X | Х | x | X | X |
| Height, weight⁵ | | x | X | | X | х | x | X | X | X | | х | x | | |
| ECG <sup>8</sup> | | X | X | | | х | X | | | | | X | | | X |
| Eliciting AEs | | x | X | X | X | X | x | X | X | X | | X | x | X | X |
| Disease Assessment and PFT | | | | | | | | | | | | | | | |
| Review SLB <sup>7</sup> (if applicable) | X | | | | | | | | | | | | | | |
| Review transbronchial lung biopsy/BAL <sup>8</sup> | | X | | | | | | | | | | | | | |
| Review HRCT <sup>7</sup> | X | | | | | | | | | | | | | | |
| HRCT | | Χ <sup>9</sup> | | | | | | | | | | X | | | X |
| Spirometry (FVC). Collection and recording of the retrospective FVC values <sup>10</sup> | | х | x | | | | | X | | | x | x | | x | x |
| Dico | | x | | | | | | | | | | | | | |
| 6MWT | | X | X | | | | | X | | | Х | Х | | X | X |
| Laboratory Tests | | | | | | | | | | | | | | | |
| Hematology, blood chemistry <sup>11</sup> | | x | X | | x | X | х | X | X | X | | X | x | X | X |
| Serologic tests <sup>11</sup> | | х | | | | | | | | | | | | | |
| Pregnancy test | | х | X <sup>12</sup> | | | X | х | X | | X | | Х | | | |
| PROs and ClinROs | | | | | | | | | | | | | | | |
| GAP assessment | | х | | | | | | | | | | | | | |



| Study period | IC<br>Visit | Screening<br>(Washout, if<br>applicable) | | Treatment period Fol | | | | | | | Follow-Up | Long-Term<br>Follow-Up <sup>16</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week<br>(Window) | | -4 to −1 | Day 1 | W1<br>(± 1 d) | W2<br>(± 2 d) | W4<br>(± 2 d) | W8<br>(± 2 d) | W12<br>(± 1 w) | W16<br>(± 1 w) | W20<br>(± 1 w) | | V26<br>1 w) | 14–28 days<br>after last<br>dose | W39<br>(± 2 w) | W52<br>(± 2 w) |
| Borg scale <sup>13</sup> | | х | х | | | | | х | | | х | х | | Х | х |
| EQ-5D questionnarie <sup>13</sup> | | х | х | | | | | х | | | | х | | | х |
| Patient diary (review, dispense) <sup>14</sup> | | | Х | х | Х | Х | Х | х | х | Х | , | Х | | · | |
| Telephone calls (IPF Care program) <sup>15</sup> | | | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup>Written informed consent must be obtained prior to any study-associated procedure, including discontinuing any prohibited medications.

<sup>&</sup>lt;sup>2</sup> Safety-related information (AEs) and adherence to treatment is collected.

<sup>&</sup>lt;sup>3</sup> Complete medical history is collected at an IC visit, washout and screening only. Thereafter, directed history (including review of AEs/SAEs, concomitant medications, oxygen use, hospitalizations, dosing, and diary) is only collected.

<sup>&</sup>lt;sup>4</sup> Complete physical examination is performed at the Screening only (head, eyes, ears, nose, and throat, and the cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, genitourinary, and neurological systems). At subsequent visits (or as clinically indicated), only limited, symptom-directed physical examinations should be performed.

<sup>&</sup>lt;sup>5</sup> Height is assessed at the Screening only.

<sup>&</sup>lt;sup>6</sup> ECG should be performed after patient's resting in a supine position for at least 10 min, prior to other procedures scheduled at that same time (e.g., vital sign measurements, blood draws), bronchodilator administration and within 3 hours after any meal)

<sup>&</sup>lt;sup>7</sup> To confirm IPF will be applicable to use previously performed HRCT, if it is performed not earlier than 24 months before the Screening. Review of the SLB samples obtained within 4 years before the Screening should be performed centrally for elig bility confirmation. Histopathological evaluation, if not available, is not repeated at the Screening.

<sup>&</sup>lt;sup>8</sup> Transbroncheal biopsy or BAL are not mandatory and will only be reviewed at the Screening, if available, to exclude other causes of PF.

<sup>&</sup>lt;sup>9</sup> HRCT should be performed at the Screening only for patients having no validated procedure within 2 months prior initiation of treatment.

<sup>&</sup>lt;sup>10</sup> At screening, spirometry measurements of FVC should be performed before and after administration of albuterol (or salbutamol) from a metered dose inhaler (4 separate doses of 100 mg). Tests should be repeated after a 15-min delay. During further visits, bronchodilator test is not necessary to perform. Collection and recording of the retrospective FVC values obtained in clinical practice over the last year will be performed only at the screening visit.

<sup>11</sup> Blood samples must be drawn in fasted state. Serologic tests: rheumatoid factor, anticyclic citrullinated peptide and antinuclear antibody titer.

<sup>12</sup> Pregnancy test must be performed before first dosing on Day 1 and must be negative. If the urine test is positive, serum pregnancy test must be performed.

<sup>&</sup>lt;sup>13</sup> Questionnaires should be self-administered before the patient or clinician receives any information on disease status, prior to the performance of non-PRO assessments, and prior to the administration of study treatment, with the exception for Borg scale administered in conjunction with the 6MWT.

<sup>&</sup>lt;sup>14</sup> Patient diary should be filled out on daily basis by the patient and reviewed by the investigator at in-clinic visits. Patient diary captures information on compliance and AEs occurance and is dispensed as needed.

<sup>&</sup>lt;sup>15</sup> Schedule of calls in IPF Care Program you can see in Appendix 7

<sup>&</sup>lt;sup>16</sup> Only in patients continuing treatment with pirfenidone in real clinical practice.

## 4.2. Randomization and Blinding<sup>2</sup>

Randomization is not planned in the study.

Blinding is not applicable in this open-label study.

## 5. Sample Size<sup>3</sup>

Taking into account study design (single group prospective study), sample size was estimated based on feasibility of patient enrollment with precision-based approach. In the ASCEND study primary efficacy endpoint (Percent Predicted FVC) in pirfenidone group changed from 67.8 (11.24) (denoted as mean (SD)) at baseline to 65.3 (14.52) at week 26, with stable disease (decline in FVC < 10 % to 0 %) in 60.1 % of study patients.

The required sample size for two-sided 95% confidence level can be calculated using the following formula:

$$\begin{split} n &= \hat{p} \hat{q} \left( \frac{Z_{\alpha/2}}{E} \right)^2; \\ n &= 0.601 \times 0.399 \left( \frac{1.96}{0.125} \right)^2 \approx 58.96. \end{split}$$

Assuming previous calculations, 60 patients included in the study will be sufficient for study parameters estimation. Taking into account study goals and the notion that the study drug is a product for the treatment of an orphan drug, margin of error of 0.125 is considered sufficient for parameter estimation. For precision-based sample size justification, with a sample size of 60 patients, an expected mean value of 2.5% and standard deviation of 20, distance from the mean to limit of the two-sided 95% confidence interval for the mean Change from Baseline to Week 26 (Percent Predicted FVC) will extend about 5 (margin of error). The SD for change from baseline at week 26 is conservatively estimated based on the results of the ASCEND study as standard deviation for Percent Predicted FVC in pirfenidone group at week 26 (14.52) multiplied by  $\sqrt{2}$  (Machin et al., 1997). This is also in line with the results of CAPACITY programme (Noble et al. 2011) in which the SD of changes from baseline was 17 - 20 at week 72.

Taking into account an expected rate of screening failures about 45%, up to 109 patients will be screened for eligibility.

#### 6. General Considerations

## 6.1. Timing of Analyses

No interim analysis is planned in this study.

<sup>&</sup>lt;sup>2</sup> This section is based on the section 4.2 "Method of treatment assignment and blinding" of clinical study Protocol.

<sup>&</sup>lt;sup>3</sup> This section is based on the section 6.1 "Determination of sample size" of clinical study Protocol.



## 6.2. Analysis Populations

The main patient samples of interest are defined as follows.

The 'All enrolled patients' set will consist of all patients who:

Gave their Informed Consent.

The 'Allocated to treatment' set will consist of all patients who:

Gave their Informed Consent and

Had successfully completed Screening procedures.

The 'Treated set' (TS) will consist of all patients who:

Were in the 'Allocated to treatment' set and

Received any dose of the study treatment.

The 'Full analysis' set (FAS) will consist of all patients who:

- Were included in the 'Treated' set and
- Had data for at least one post-baseline assessment of any efficacy measurement.

The 'Complete case set' (CCS) will include FAS patients who

• Provided FVC data at 26-week assessment.

## 6.3. Missing Data<sup>4</sup>

For missing FVC data imputation, patients will be classified into different patterns depending on the availability of data:

Patients with a 26 week FVC value:

- 1. those who received study drug until 26 weeks (completed the treatment period);
- 2. those who prematurely discontinued study drug, but who were followed up until Week 26.

Patients without a 26 Week FVC value:

- 3. those who were alive at 26 weeks;
- 4. those who died before 26 weeks.

Missing data at other visits before Week 26 (primary outcome variable) will not be imputed. The following imputation methods including sensitivity analyses will be applied for patients with pattern 3 - 4:

Assuming that deaths of the patients (pattern 4) is likely to be related to worsening of IPF, these unobserved FVC values should be lower than those in patients who did not die prior to Week 26. Methods for handling missing data due to death will include the following:

- Replacement with the worst possible value (FVC= 0 mL or 0%) (Primary analysis).
- Replacement with worst observed averaged FVC value at week 26 (Sensitivity analysis).

<sup>&</sup>lt;sup>4</sup> This section is based on the section 6.2 "Summaries of conduct of study" of clinical study Protocol.



• Replacement with an intermediate value (FVC =1500 mL or 50%) (Sensitivity analysis).

Missing data due to reasons other than death (e.g., missing visits, early withdrawal from the study, including missing values due to lung transplantations) (pattern 3) will be replaced with imputed values based on the average measurements for "similar" patients at that time point. Similar patients are those without missing data before that time point and whose data have the smallest sum of squared deviations (SSD) from that patient for all visits prior to the one with the missing data. Missing data due to lung transplant will be imputed using the SSD method even if the patient dies after lung transplant.

The procedure referred to as the sum of squared deviations (SSD) is outlined as follows:

**Step 1:** For post-Baseline missing value to be imputed at a visit (Visit week 26) for a particular patient (Patient A), a set of all patients without any missing values for visits from Baseline up to Visit week 26 as Patient A will be selected.

**Step 2:** For the patients in this set, the SSDs between each patient selected in Step 1 and Patient A will be calculated across all non-missing values from Baseline up to the visit prior to Visit week 26.

**Step 3:** The 3 patients with the smallest SSDs will be identified and the average of their non-missing value at Visit week 26 will be used to impute the missing value for Patient A at that visit. The number of smallest SSDs to calculate the average can be less than 3 due to availability of patients defined in Step 1 or more than 3 based on tied SSDs.

A sensitivity analysis will use the data imputed with last observation carried forward method (LOCF).

Complete case analysis will also be performed as a sensitivity analysis.

If the information about end date for prior/concomitant therapy is missing or incomplete, the following rules (table 6.1) will be used for the classification of therapy as prior or concomitant.

Table 6.1 – Management of partial and missing prior/concomitant therapy end date.

| Day | Month | Year | Processing |
|---|---|---|---|
| is missing | is known | is known | Therapy will be classified as concomitant, if month and year ≥ month and year of the first dose of study |
| is missing | is missing | is known | therapy, else – as prior Therapy will be classified as |
| is known | is missing | is known | concomitant, if year ≥ year of the first dose of study therapy, else – as prior |
| is missing | is known | is missing | |
| is known | is known is missing | | Therapy will be classified as concomitant |
| is missing | is missing | is missing | Conconntant |



If the information about adverse event start date and time is missing or incomplete, the following rules (table 6.2) will be used for the classification of adverse events as TEAEs and non-TEAEs (occurred before the start of study treatment).

Table 6.2 – Management of partial and missing AE start date.

| Day | Month | Year | Processing |
|---|---|---|---|
| | | | AE will be classified as TEAE, if month |
| is missing | is known | is known | and year $\geq$ month and year of the first |
| | | | dose of study therapy |
| is missing | is missing | is known | AE will be classified as TEAE, if year ≥ |
| is known | is missing | is known | year of the first dose of study therapy |
| is missing | is known | is missing | AE will be classified as |
| is known | is missing | is missing | TEAE |
| is missing | is missing | is missing | IEAE |

No date imputation will be performed for listings.

## 6.4. Interim Analyses and Data Monitoring<sup>5</sup>

No interim analysis is planned in the study.

#### 6.5. Multi-center Studies

Data from all centers will be merged and analyzed as one population for all study endpoints.

## 6.6. Multiple Testing

No adjustment for multiplicity is planned.

#### 7. Summary of Study Data

Demographic and other baseline characteristics, efficacy and safety data will be summarized by time point of assessment and listed.

#### **Default Summary Statistics**

The default summary statistics for quantitative and ordinal variables will be the number of observations (n), mean, standard deviation (SD), median, minimum (Min) and maximum (Max).

#### **Default Frequency Tabulations**

For qualitative variables, the number and percentage (n, %) of patients with non-missing data per category and total number of patients with non-missing data where applicable (n') will be the default summary presentation.

For AEs and medical history, however, the denominator for the percentage calculation will be the number of patients at risk. A patient will be considered at risk if the patient is in the Treated set.

<sup>&</sup>lt;sup>5</sup> This section is based on the section 6.6 "Interim analysis" of clinical study Protocol.



The number of decimals for each descriptive statistic will be determined by the following rules:

- mean, median: +1 decimal symbols compared to the analysed variable values;
- standard deviation: +2 decimal symbols compared to the analysed variable values;
- minimum and maximum values: the same as for the analysed variable values;
- percentages will be rounded to one decimal symbol;
- confidence intervals will be presented with accuracy of the estimated value.

The maximum number of decimal places in the statistical report is four. If some descriptive statistic has more than four decimal places after above mentioned rules application, this value will be rounded to four decimal places.

#### Statistical Tests and Common Calculations

Unless otherwise specified in the description of the analyses, the following arrangements will be applied:

- 95% two-sided confidence intervals (CI);
- [if appropriate] CIs for mean values will be calculated based on normal distribution (SAS procedure UNIVARIATE with CIBASIC option);
- [if appropriate] CIs for proportions will be computed using the exact (Clopper-Pearson) method.
- Type I error values (p-values) will be rounded to four decimal symbols.

For descriptive statistics and analysis, the following rules will be applied:

"<XX" results (e.g. below the limit of quantification, BLQ) will be replaced by the "XX/2" values;</li>

For quantitative measurements, changes from baseline will be calculated as [value at post-baseline visit X – baseline value].

For change from baseline, the baseline value for a variable in common cases (except for efficacy analysis) is defined as the last non-missing value collected before the first study drug administration.

Study day for each event will be calculated from the reference start date (date when patient was first exposed to study drug).

If the date of the event is on or after the reference date, then

$$study day = (date \ of \ event - reference \ date) + 1.$$

If the date of the event is prior to the reference date, then

$$study day = (date of event - reference date).$$

For partial dates study day will not be calculated.

The following visit windows will be defined:



| Visit | First day of the visit window | Last day of the visit window |
|---|---|---|
| Week 1 Telephone Assessment (+/- 1 day) | 1 | 8 |
| Week 2 (+/- 2 days) | 6 | 16 |
| Week 4 (+/- 2 days) | 20 | 30 |
| Week 8 (+/- 2 days) | 48 | 58 |
| Week 12 (+/- 2 days) | 76 | 86 |
| Week 16 (+/- 1 week) | 99 | 119 |
| Week 20 (+/- 1 week) | 127 | 147 |
| 1st day at Week 26 (+/- 1 week) | 169 | 189 |
| 2nd day at Week 26 (+/- 1 week) | 169 | 189 |
| Week 39 (+/- 2 weeks) | 253 | 287 |
| Week 52 (+/- 2 weeks) | 344 | 378 |

The data from all subjects who were treated in the rollover study will be pulled for the analysis irrespective of the trade name(s) of pirfenidone used by the subject (Esbriet® or other, if applicable). An explanatory footnote will be added to the outputs where necessary to indicate which pharmaceutical product was used.

#### 7.1. Subject Disposition

The following patient disposition summaries will be provided:

- A summary of the number of patients signed the Informed Consent and the number of screen failures with reasons for premature study termination
- A summary of the number of screen failure patients violated any inclusion/exclusion criterion, by criterion
- A summary of the number of patients allocated to treatment, the number and percentage of treated patients, the number and percentage of patients attended each study visit, the number and percentage of patients who were included into rollover study (Allocated to treatment set)
- A summary of the number and percentage of patients included in each population for statistical analysis (Allocated to treatment set)
- A summary of the number and percentage of patients completed the study and prematurely discontinued from the study by major reason for discontinuation (Allocated to treatment set).

By-patient listings of disposition details will be provided for all patients who signed the Informed Consent.

#### 7.2. Protocol Deviations<sup>6</sup>

Number and percentage of patients with at least one protocol deviation will be tabulated (Allocated to treatment set). All protocol deviations will be listed (All Enrolled patients).

\_

<sup>&</sup>lt;sup>6</sup> This section is based on the section 9.2 "Protocol deviations" of clinical study Protocol.



#### 7.3. Demographic and Baseline Variables 7

eCRF form: "DEMOGRAPHIC DATA", "VITAL SIGNS".

Descriptive statistics for the following demographic and anthropometric characteristics, which are evaluated at screening, will be presented in accordance with section 7:

- demographic characteristics: age, gender, race, ethnicity;
- anthropometric characteristics: height (cm), weight (kg), body mass index (BMI, kg/m<sup>2</sup>).

Body mass index will be calculated as weight  $(kg) / [height (m)]^2$ .

eCRF form: "SURGICAL LUNG BIOPSY", "REVIEW TRANSBRONCHIAL LUNG BIOPSY/BAL", "HRCT SCAN FOR PATIENT ELIGIBILITY CONFIRMATION", "DL(CO)", "SPIROMETRY", "SEROLOGIC TESTS", "GAP RISK ASSESSMENT".

The following parameters will be tabulated in accordance with section 7:

- Disease Assessment and PFT:
  - Surgical lung biopsy (SLB) (if available) (UIP pattern assessment of regional specialist: Consistent, Probable, Possible, Inconsistent / unclassified; UIP pattern assessment of central specialist: Consistent, Probable, Possible, Inconsistent / unclassified)
  - o Transbronchial lung biopsy/ Bronchoalveolar lavage (BAL) (if available) (Are there features supporting an alternative diagnosis? Yes/No)
  - High-resolution computed tomography (HRCT) (HRCT fibrosis score; Lung opacity score (Ground-glass opacity ))
  - HRCT scan for patient's eligibility confirmation (UIP pattern assessment of regional CT-specialist: Typical (apparent), Possible; UIP pattern assessment of central CT-specialist: Typical (apparent), Possible, Inconsistent)
  - Carbon monoxide diffusing capacity (DL<sub>CO</sub> predicted)
  - Pre-, post- bronchodilator, and retrospective FVC (absolute), ml; FVC (relative),
     predicted, pre- post-bronchodilator FEV1/FVC,
- Laboratory Tests:
  - Serologic tests: rheumatoid factor, anticyclic citrullinated peptide and antinuclear antibody titer (Positive / Negative)
- PROs and ClinROs:
  - GAP (Gender, Age, Physiology) assessment (Stage, GAP Index (Points), Mortality 1-yr, Mortality 2-yr, Mortality 3-yr)

Specific calculations and/or conversions include but are not limited to the following:

**DL**<sub>CO</sub>: Data for DL<sub>CO</sub> will be collected in the eCRF. Results of DL<sub>CO</sub> measurements will be corrected to patients' hemoglobin (Hb) using one of the formulas (Cotes et al. 1979):

Hb-corrected DL<sub>CO</sub> for men: DL<sub>CO</sub> ×  $(10.22 + \text{Hb})/(1.7 \times \text{Hb})$ 

CONFIDENTIAL AND PROPRIETARY Data MATRIX Ltd.

<sup>&</sup>lt;sup>7</sup> This section is based on the section 6.3 "Summaries of Demographic and Baseline characteristics", 4.5.6 "HRCT and Surgical Lung Biopsy", 4.5.7 "Spirometry and DL<sub>CO</sub> Measurements", 4.5.8 "Laboratory, Biomarker, and Other Biological Samples", 4.5.11.4 "GAP Risk Assessment System" of clinical study Protocol.



Hb-corrected DL<sub>CO</sub> for women: DL<sub>CO</sub> ×  $(9.38 + Hb)/(1.7 \times Hb)$ 

where Hb indicates the value of hemoglobin, in g/dL. If the Hb value is reported in g/L, then the Hb value is divided by 10. If the Hb value is reported in mmol/L, then the Hb value is divided by 0.6206.

Use the hemoglobin value available on the same day if possible; otherwise, the closest hemoglobin value before or after the actual  $DL_{CO}$  assessment date should be used. If the two values are equidistant, the value before the actual  $DL_{CO}$  assessment should be used.

All data will be listed.

#### 7.4. Concurrent Illnesses and Medical Conditions<sup>8</sup>

eCRF form: "GENERAL MEDICAL HISTORY", "HISTORY OF IDIOPATHIC PULMONARY FIBROSIS".

Medical history findings will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 22.0 (or further updating) according to Data MATRIX SOP [4], and will be presented by Primary System Organ Class (SOC) and Preferred Term (PT) within SOC.

Medical history events marked as "Resolved" will be considered as prior diseases. Medical history events marked as "Ongoing" will be considered as concomitant diseases.

Prior and concomitant diseases will be tabulated separately.

Medical history findings will be reported on a by-patient basis. This implies that if the patient suffered the same event (mapped to same PT) repeatedly the event will be counted once and only once for appropriate SOC. Within SOC patients may have reported more than one PT. The SOCs and PTs within each SOC will be sorted by descending order of total incidence.

As medical history of main disease, the following parameters: (Idiophatic Pulmonary Fibrosis), Duration of clinical symptoms consistent with IPF (months), Clinically significant environmental exposure known to cause pulmonary fibrosis (Yes/ No), Known explanation for interstitial lung disease (Yes/ No), Cigarette smoking within 28 days before the treatment start (Yes/ No) will be presented descriptively in the separate table.

All data will be listed.

#### 7.5. Prior and Concurrent Medications<sup>9</sup>

eCRF form: "PRIOR/ CONCOMITANT MEDICATIONS".

CONFIDENTIAL AND PROPRIETARY Data MATRIX Ltd.

<sup>&</sup>lt;sup>8</sup> This section is based on the section 4.5.2 "Medical History and Demographic Data", 6.3 "Summaries of Demographic and Baseline characteristics" of clinical study Protocol.

<sup>&</sup>lt;sup>9</sup> This section is based on the section 6.2 "Summaries of conduct of study" of clinical study Protocol.



- 1. Prior and concomitant medications will be analyzed based on the information from the Concomitant/Prior Medications (CM) domain.
- 2. All prior and concomitant medications will coded using the World Health Organization Drug Dictionary (WHODD) version B2 March 2018 (or further updating) according to Data MATRIX SOP [4].

Classification of treatment as either Prior or Concomitant will be based on stop date of medication in "PRIOR/CONCOMITANT" eCRF form. The number (%) of patients reporting the use of any medications, and the number of reported medications will be presented in separate tables by pharmacological subgroup (3rd level) and chemical substance (5th level).

Medications that stop prior to the date of first dose of study therapy will be classified as Prior medications. If a medication stops on or after the date of first dose of study therapy (or "ONGOING") then the medication will be classified as Concomitant. For patients who take part in the rollover study, medications started on or after the date of the first dose of the study drug during the rollover study will be summarized separately.

3. If the information about stop date of medication is missing or incomplete, the rules from section 6.3 will be applied for classification. Medications will be assumed to be concomitant, unless there is clear evidence (through comparison of partial dates) to suggest that the medication stopped prior to the first dose of study therapy. If there is clear evidence to suggest that the medication stopped prior to the first dose of study therapy, the medication will be assumed to be Prior.

By-patient listings will be provided.

## 8. Efficacy Analyses<sup>10</sup>

eCRF form: "SPIROMETRY".

Descriptive statistics for all efficacy variables will be presented by visit. For the descriptive statistics, the rules presented in section 7 will be applied.

The FAS and Complete case set will be used for the efficacy analysis. Analysis on Complete case set will be one of the sensitivity analyses to be performed.

All efficacy data will be listed.

#### 8.1. Primary Efficacy Analysis

The primary outcome variable is the absolute change in FVC from Baseline to Week 26 (both in mL and % predicted). Baseline FVC will be the average of the FVC measured at the Screening (excluding values after bronchodilator administration) and Day 1 visits, if either is missing, the non-missing value will be used. The FVC at Week 26 will be the average of the FVC measured on

\_

<sup>&</sup>lt;sup>10</sup> This section is based on the section 6.4 "Efficacy analyses" of clinical study Protocol.



two separate days at Week 26, if either is missing, the non-missing value will be used. If both values are missing, the data will be imputed as specified in Section 6.3.

Data will be analyzed using standard descriptive statistics for continuous variables and 95% CI for the means and mean changes.

The data imputation methods for primary endpoint are described in Section 6.3.

For the primary analysis, missing data due to death will be replaced with the worst possible value (FVC= 0 mL or 0%). Missing data due to reasons other than death (pattern 3) will be replaced with imputed values based on the average measurements for "similar" patients at that time point (SSD, Primary analysis).

As sensitivity analyses, the following imputation methods will be used:

- 1. Missing data due to death will be replaced with the worst observed FVC value at week 26. Missing data due to reasons other than death (pattern 3) will be replaced with imputed values based on the average measurements for "similar" patients at that time point (SSD).
- 2. Missing data due to death will be replaced with an intermediate value (FVC =1500 mL or 50%). Missing data due to reasons other than death (pattern 3) will be replaced with imputed values based on the average measurements for "similar" patients at that time point (SSD).
- 3. Missing data due to death will be replaced with the worst possible value (FVC= 0 mL or 0%). Missing data due to reasons other than death (pattern 3) will be replaced with LOCF.
- 4. Missing data due to death will be replaced with the worst observed FVC value at week 26. Missing data due to reasons other than death (pattern 3) will be replaced with LOCF.
- 5. Missing data due to death will be replaced with an intermediate value (FVC =1500 mL or 50%). Missing data due to reasons other than death (pattern 3) will be replaced with LOCF.
- 6. Missing data due to death and due to reasons other than death (pattern 3) will be replaced with LOCF.

Analysis of the primary efficacy endpoint will be also repeated on the Complete case set (CCS) without missing data imputation as the sensitivity analysis. Complete case set will include patients related to pattern 1 and 2 (section 6.3), results will be reported for pattern 1 and 2 separately and overall.

Primary analysis with missing data imputation of the primary efficacy endpoint and analysis on the CCS set will also be repeated excluding all values outside of visit window based on visit window definitions in Section 7.

For this analysis, if one of the observations pertaining to Week 26 visit is within the visit window and the other is outside the visit window, the observation which is within the visit window will be used for Week 26 assessment. The distribution (number and percentage) of primary outcome variable across three categories of change from Baseline (Decline of  $\geq 10\%$  or death



before Week 26; Decline of < 10% to 0%; Improvement of  $\geq$  0%) (absolute change in FVC % predicted and relative change for volume) will be provided in frequency table.

Additionally, the absolute change in FVC from Baseline at Week 12, 39 (optional) and 52 (optional) and mean FVC values through all time points (both in mL and % predicted) will be summarized (without missing value imputation) in tables with standard descriptive statistics for continuous variables and 95% CI for the means and mean changes. For each time point, descriptive analysis will be repeated for values within visit window.

#### 8.2. Secondary Efficacy Analyses

eCRF form: "6-Minute Walk Test", "BORG SCALE", "EUROPEAN QUALITY OF LIFE 5-DIMENSION 5-LEVEL QUESTIONNAIRE".

## Change in 6MWT distance from Baseline to Week 26

Baseline 6MWT distance will be the average of the measurements recorded at the Screening and Day 1 visits. The 6MWT distance at Week 26 will be defined as the average of the 6MWT distance recorded on two separate days at Week 26. Data will be analyzed using standard descriptive statistics for continuous variables and 95% CI for the means and mean absolute changes.

The distribution (number and percentage) of 6MWT distance across three categories of change from Baseline (Decline of  $\geq 50$  m or death before Week 26; Decline of  $\leq 50$  m to 0 m (exclusively), Improvement of  $\geq 0$  m) will be provided in frequency table.

Additionally, the absolute change in 6MWT from Baseline at Week 39 (optional) and Week 52 (optional) will be summarized in table with standard descriptive statistics for continuous variables and 95% CI for the mean.

Borg scale results will be presented descriptively by visit of assessment. Borg scale results (as a continuous variable) will be presented for both pre-test and post-test by visit of assessment and change from baseline (the average of the measurements recorded at the Screening and Day 1 visits) at post-baseline visits for pre-test assessments only.

The Borg scale results at Week 26 will be defined as the average of the Borg scale results recorded on two separate days at Week 26. If at baseline and/or at Week 26 for 6MWT distance or Borg scale either value is missing, the non-missing value will be used.

Descriptive analysis for 6MWT distance and Borg scale results will be repeated excluding assessments outside of visit window.

## Change from Baseline to Week 26 in patients' quality of life as measured with EQ-5D-5L

• Cross tabulation for each of five dimensions (Mobility, Self-Care, Usual Activities, Pain / Discomfort, Anxiety / Depression) by response and study week.



- VAS score, including absolute changes from baseline, will be summarized with descriptive statistics by study week.
- EQ-5D-5L index score using the UK value set, including absolute changes from baseline, will be summarized with descriptive statistics by study week.

Descriptive analysis will be repeated excluding assessments outside of visit window.

The baseline assessment is the last non-missing assessment prior to the first dose of the study drug.

## 8.3. Exploratory Efficacy Analyses

eCRF form: "HRCT SCAN", "ADVERSE EVENTS".

#### HRCT fibrosis score

The HRCT findings will be evaluated using HRCT scoring system. One ILD radiologist will make assessments of 4 main findings in three zones of each lung. The six zone scores will be averaged to determine the total score for each patient. Score will be recorded at the initial diagnosis and after six and 12 months in a similar manner for further comparison. The mean  $\pm$  SD of HRCT fibrosis score like continuous variable will be determined obligatory at baseline, 6 months and optional at 12 months.

The values of HRCT fibrosis score at baseline, at Week 26 and Week 52 (optional) will be summarized in table with standard descriptive statistics for continuous variables and 95% CI for the mean.

Additionally, the absolute change of HRCT fibrosis score from baseline at Week 26 and Week 52 (optional) will be summarized in table with standard descriptive statistics for continuous variables and 95% CI for the mean.

The paired t-test will be performed to evaluate the changes in the variable from the baseline to Week 26 and Week 52 (optional), respectively. The type I error rate will be set to 5%.

## Lung opacity (ground-glass attenuation)

The sign 'lung opacity' will be qualified separately using methodology described above for other signs, and its change over time will be assessed outside the framework of a total summed index of fibrosis (HRCT fibrosis score). Lung opacity should be graded as reticular abnormality to calculate the score for each zone, i.e. the percentage (%) area of opacity in a zone should be multiplied by the score of 2.

The lung opacity score at Baseline, at Week 26 and Week 52 (optional) will be summarized using standard descriptive statistics for continuous variables and 95% CI for the mean.

Additionally, the absolute change of lung opacity score from Baseline at Week 26 and Week 52 (optional) will be summarized in table with standard descriptive statistics for continuous variables and 95% CI for the mean.



#### Exacerbations

An exacerbation will be defined as an AE with special criteria "Is this an exacerbation of IPF?" = "Yes", i.e. only in case the exacerbation has led to death of a patient. Rate of exacerbation will be reported in three following tables:

- Exacerbation cases during treatment period (until Week 26).
- Exacerbation cases during long-term follow-up period (from Week 26 to Week 52).
- Exacerbation cases during whole study period (from Day 1 to Week 52, applicable only for patients continuing in the rollover study).

Exacerbation cases will be listed.

The treatment period and rollover period for the analysis of exacerbations will be defined similarly to Section 9.2.

#### 9. Safety Analyses

#### 9.1. Exposure

Exposure will be evaluated based on the information from the "ASSESSMENT OF COMPLIANCE", "STUDY DRUG ADMINISTRATION (TREATMENT PERIOD)", "COMMERCIALLY AVAILABLE PIRFENIDONE ADMINISTRATION (ROLLOVER STUDY)" eCRF form.

Pirfenidone will be taken orally in a daily dose of 2403 mg in divided doses three times per day with food. Study treatment should be titrated over 14 days, as tolerated, to the full dose of 9 capsules per day (three capsules TID), as follows:

- Days 1 to 7: one capsule TID (801 mg/day)
- Days 8 to 14: two capsules TID (1602 mg/day)
- Day 15 and continuing: three capsules TID (maximum of 9 capsules daily equal to 2403 mg/day).

Study treatment will continue until visit at Week 26 ( $\pm$  1 week), unless terminated earlier for reasons described in Section 4.6.2 of the Protocol or patient is proceeding in the rollover study.

The total duration of exposure is defined as the time interval in weeks between the first dose and the last dose, inclusive, of study drug based on the patient study drug dosing information. Total duration (weeks) of exposure to study drug in the Treated set will be summarized by study period using descriptive statistics.

Exposure (duration of therapy during rollover study and overall up to 58 weeks) for patients in the rollover study will also be presented descriptively.



Descriptive statistics for Total number of capsules taken during the study period will also be presented.

All exposure data will be listed.

#### 9.2. Adverse Events

eCRF form: "ADVERSE EVENTS".

AEs will be reported on a per-patient basis, i.e. counting patients rather than events.

After informed consent has been obtained but prior to initiation of study drug, only serious adverse events caused by a protocol-mandated intervention should be reported.

After initiation of study drug, all adverse events will be reported until 28 days after the last dose of study drug. Additionally, for patients continuing in the rollover part of the study adverse events will be reported until Week 52.

Only treatment emergent AEs will be summarized. In the listings, however, all occurrences of the AEs will be presented. Treatment emergent AEs will be summarized per primary SOC and PT. Severity of treatment emergent AEs will be summarized separately.

Treatment-emergent AE is any reported adverse event that starts after initiation of the study therapy and up to 28 days after the last dose of study therapy.

All registered AEs will be coded using the MedDRA version 22.0 (or further updating) and tabulated in the report with grouping by primary system organ class (SOC) and preferred term (PT).

Number (percentage) of patients and number of AEs will be presented for the Treated Set in the following tables:

- All treatment-emergent AE / SAE;
- Treatment-emergent AE / SAE related to the study drug ("Is the adverse event suspected to be caused by the study drug on the basis of facts, evidence, science-based rationales, and clinical judgment?" = "Yes" including those events where assessment is missing);
- TEAE by maximum severity (Severity, CTCAE v.4.0);
- TEAE related to study drug by maximum severity (Severity, CTCAE v.4.0);
- TEAE leading to the permanent discontinuation of study drug (Action taken with IMP="Permanently discontinued");
- TEAE leading to death (AE with Outcome = "Death") including TEAE related to the study drug;
- TEAE related to the study drug leading to death;
- TEAE of special interest ("Is this an adverse event of special interest?" = "Yes");
- Non-serious TEAEs that occurred at a frequency of >= 5% (if no events occurred at the 5% threshold all non-serious TEAEs will be tabulated).



This set of tables will be repeated for the following study periods:

- Treatment period defined as first dose of study drug to last dose of study drug in the treatment period + 28 days or until the first dose in the rollover period (Treated Set).
- Rollover period defined as first dose in the rollover to last dose in the rollover study + 28 days (Treated Set, patient continuing in the rollover study).

Tables of TEAEs by maximum severity will be prepared using the following rules: each SOC / PT category will include only the AEs with the worst severity for each patient. In the Overall category, all AEs of the patient will be presented. Each patient will be counted only once with the worst severity in each SOC and each PT level as well as in the Overall level.

Number of patients who died will be tabulated.

All AEs/SAEs will be listed. Non-treatment emergent adverse events will be identified accordingly in the listing.

#### 9.3. Pregnancies

eCRF form: "URINE PREGNANCY TEST".

All women of childbearing potential will have a urine pregnancy test at the Screening and on Day 1 before start of treatment. Urine pregnancy tests will be performed repeatedly at specified subsequent visits as scheduled in the Table 1.

The results of these tests and pregnancies episodes will be reported in the listing.

## 9.4. Clinical Laboratory Evaluations

eCRF form: "HEMATOLOGY", "SERUM CHEMISTRY".

Clinical laboratory evaluations as scheduled in the Table 1 include the following parameters:

- hematology (plasma): white blood cells (WBC) count, red blood cells (RBC) count, hemoglobin, hematocrit, platelet count, (relative) differential WBC count (neutrophils, eosinophils, basophils, monocytes, lymphocytes);
- blood chemistry panel (serum or plasma): albumin, alkaline phosphatase (AP), ALT, AST, direct bilirubin, total bilirubin, total protein, cholesterol, creatine kinase (CK), creatinine, triglycerides, gamma-glutamyl transferase (GGT), glucose, lactic dehydrogenase (LDH), calcium, phosphorus, magnesium, potassium, sodium, urea nitrogen, uric acid;

Creatinine clearance should be assessed at the Screening for eligibility confirmation using the following formula by Cockcroft-Gault (Cockcroft DW et al, 1976):

For serum creatinine concentration in mg/dL:



 $CrCl (mL/min) = (140 - age (years)) \times weight (kg) \times 1.0 / 72 \times serum creatinine (mg/dL)$ 

For serum creatinine concentration in µmol/L:

CrCl (mL/min) =  $(140 - age (years)) \times weight (kg) \times 1.0 / 0.81 \times serum creatinine (\mu mol/L)$ 

For laboratory parameters the following tables will be presented according to section 7:

- descriptive statistics of measured values and changes from baseline (including creatinine clearance);
- shift tables based on comparison with normal range (Lower/Normal/Higher);
- frequency tables for Out of range: No/Yes clinically significant (Yes CS) / Yes nonclinically significant (Yes NCS) for laboratory parameters.

All laboratory data will be listed.

## 9.5. Other Safety Measures

eCRF form: "VITAL SIGNS", "ECG", "PHYSICAL EXAMINATION".

#### Vital signs

Vital signs (respiratory rate (breaths/ minute), pulse rate (beats/ minute), and systolic and diastolic blood pressure (mmHg), and axillary temperature (°C)), body weight (kg) and body height (cm) results will be presented in accordance with section 7.

Vital signs results will be presented by visit of assessment as scheduled in the Table 1. Body height will be assessed only at screening.

Vital signs and body weight results will be presented as the following outputs:

- descriptive statistics for measured values and changes from baseline (vital signs, body weight, BMI);
- frequency tables for Out of range: No/Yes clinically significant (Yes CS) / Yes non-clinically significant (Yes NCS) (vital signs).

All data will be listed.

#### **ECG**

A 12-lead electrocardiogram (ECG) results will be represented in accordance with section 7 by visit of assessment as scheduled in the Table 1 as the following outputs:

 shift table by post baseline visit compared to baseline for Normal/Abnormal clinically significant (Abnormal CS) / Abnormal non-clinically significant (Abnormal NCS) evaluation for General assessment



- descriptive statistics of ECG parameters and their changes from baseline (Heart rate, beats/min; QT interval, ms; QTC-F interval, ms).
- frequency table for Out of range: No/Yes clinically significant (Yes CS) / Yes non-clinically significant (Yes NCS) for ECG parameters.

All ECG data will be listed.

## Physical examinations

Complete physical examination is performed at the Screening only (head, eyes, ears, nose, and throat, and the cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, genitourinary, and neurological systems). At subsequent visits, only limited, symptom-directed physical examinations should be performed.

Physical examination results as scheduled in the Table 1 will be presented in accordance with section 7 by visit of assessment as the following output:

frequency table for Normal/Abnormal clinically significant (Abnormal CS) / Abnormal non-clinically significant (Abnormal NCS) evaluation.

All physical examination data will be listed.

#### 10. Pharmacokinetics

Not Applicable.

#### 11. Other Analyses

Not Applicable.

#### 12. Reporting Conventions

Not Applicable.

#### 13. Technical Details

Statistical analysis will be performed using SAS 9.4.

One (final) statistical analysis report will be prepared in the Microsoft Office Word (.docx) format after the end of data collection and database lock. The results of statistical analysis will be presented in the form of tables, figures and listings in English.

#### 14. Summary of Changes to the Protocol



The analyses methods in this SAP are fully consistent with the clinical study Protocol.



#### 15. References

- 1) Committee for Proprietary Medicinal Products (CPMP). International Conference on Harmonisation (ICH) Topic E9: Note for Guidance on Statistical Principles for Clinical Trials; September 1998.
  - 2) DataMatrix SOP STAT001 Statistical Principles ver.3.0 June 2019.
- 3) DataMatrix\_SOP\_STAT002\_Statistical Analysis Plan Development\_ver.2.0\_July 2017.
- 4) DataMatrix\_SOP\_DM010\_Dictionary Management and Data Coding ver.2.0 August 2015.
- 5) Machin D., Campbell M., Fayers P., Pinol A. "Sample size tables for clinical studies"// Second edition Blackwell Science Ltd, 1997.
- 6) Noble PW, Albera C, Bradford WZ et al. CAPACITY Study Group. Pirfenidone in patients with idiopathic pulmonary fibrosis (CAPACITY): two randomised trials. Lancet 2011, 377:1760–1769.
  - 7) ML39355 Study Results Posting Requirements.



#### 16. Listing of Tables, Listings and Figures

#### 16.1. Tables

## Patients Disposition

Table 1.1 Patients disposition (All Enrolled patients)

Table 1.2 Violation of eligibility criteria (Screening Failures)

Table 1.3 Analysis populations (Allocated to treatment set)

Table 1.4 Study visits

#### **Protocol Deviations**

Table 1.5 Protocol deviations / violations (Allocated to treatment set)

#### Demographic and Anthropometric characteristics

Table 1.6 Demographic characteristics (TS)

Table 1.7 Anthropometric characteristics (TS)

#### Baseline Variables

Table 1.8 Surgical lung biopsy (TS)

Table 1.9 HRCT for patient eligibility confirmation (TS)

Table 1.10 Carbon monoxide diffusing capacity (DLCO) (TS)

Table 1.11 Pre- and post-bronchodilator spirometry parameters at screening (TS)

Table 1.12 Serologic tests (TS)

Table 1.13 GAP assessment (TS)

Table 1.14 Review transbronchial lung biopsy/BAL (TS)

#### Medical history

Table 1.15 Prior medical/surgical conditions/diagnoses (TS)

Table 1.16 Concurrent medical/surgical conditions/diagnoses (TS)

Table 1.17 History of idiopathic pulmonary fibrosis (TS)

#### Prior and concomitant medications

Table 1.18 Prior medications (TS)

Table 1.19 Concomitant medications (TS)

Table 1.20 Concomitant medications during rollover study (TS)

#### Efficacy Analyses

Table 2.1 Descriptive statistics for FVC by visit (FAS)

Table 2.2 Primary efficacy endpoint (FAS)

Table 2.3 Primary efficacy endpoint: categorical results (FAS)

Table 2.4 Primary efficacy endpoint by pattern type (CSS)

Table 2.5 6-Minute Walk Test (FAS)

Table 2.6 Change in 6MWT distance at Week 26 by category (FAS)

Table 2.7 Borg scale (FAS)

Table 2.8 EQ-5D-5L. Descriptive statistics (FAS)

Table 2.9 Change in EQ-5D-5L. Mobility (FAS)

Table 2.10 Change in EQ-5D-5L. Self-Care (FAS)

Table 2.11 Change in EQ-5D-5L. Usual Activities (FAS) Table 2.12 Change in EQ-5D-5L. Pain/Discomfort (FAS)

Table 2.13 Change in EQ-5D-5L. Anxiety/Depression (FAS)

Table 2.14 EQ-5D-5L. VAS and Index score (FAS)

Table 2.15 HRCT. HRCT fibrosis score (FAS)

Table 2.16 HRCT. Lung opacity score (FAS)

Table 2.17 Exacerbation cases during treatment period (FAS)  $\,$ 

Table 2.18 Exacerbation cases during rollover study (FAS, patients continuing in the rollover study)

Table 2.19 Exacerbation cases during whole study period (FAS, patients continuing in the rollover study)

#### Safety Analyses

Table 3.1 Duration of exposure (TS)

Table 3.2 Total number of capsules taken (TS)

Table 3.3.1 Treatment-emergent adverse events during treatment period (TS)

Table 3.3.2 Treatment-emergent adverse events during rollover study (TS, patients continuing in the rollover study)

Table 3.3.3 Treatment-emergent adverse events during whole study period (TS)

Table 3.4.1 Treatment-emergent adverse events related to the study drug during treatment period (TS)

Table 3.4.2 Treatment-emergent adverse events related to the study drug during rollover study (TS, patients continuing in the rollover study)



- Table 3.4.3 Treatment-emergent adverse events related to the study drug during whole study period (TS)
- Table 3.5.1 Serious treatment-emergent adverse events during treatment period (TS)
- Table 3.5.2 Serious treatment-emergent adverse events during rollover study (TS, patients continuing in the rollover study)
- Table 3.5.3 Serious treatment-emergent adverse events during whole study period (TS)
- Table 3.6.1 Serious treatment-emergent adverse events related to the study drug during treatment period (TS)
  - Table 3.6.2 Serious treatment-emergent adverse events related to the study drug during rollover study (TS, patients continuing in the rollover study)
  - Table 3.6.3 Serious treatment-emergent adverse events related to the study drug during whole study period (TS)
- Table 3.7.1 Treatment-emergent adverse events during treatment period by maximum severity (TS)
- Table 3.7.2 Treatment-emergent adverse events during rollover study by maximum severity (TS, patients continuing in the rollover study)
  - Table 3.7.3 Treatment-emergent adverse events during whole study period by maximum severity (TS)
- Table 3.8.1 Treatment-emergent adverse events related to the study drug during treatment period by maximum severity (TS)
  - Table 3.8.2 Treatment-emergent adverse events related to the study drug during rollover study by maximum severity (TS, patients continuing in the rollover study)
  - Table 3.8.3 Treatment-emergent adverse events related to the study drug during whole study period by maximum severity (TS)
- Table 3.9.1 Treatment-emergent adverse events of special interest during treatment period
- Table 3.9.2 Treatment-emergent adverse events of special interest during rollover study (TS, patients continuing in the rollover study)
  - Table 3.9.3 Treatment-emergent adverse events of special interest during whole study period (TS)
- Table 3.10.1 Treatment-emergent adverse events leading to death during treatment period
- (TS) Table 3.10.2 Treatment-emergent adverse events leading to death during rollover study (TS,  $\alpha$ )
  - patients continuing in the rollover study)
    Table 3.10.3 Treatment-emergent adverse events leading to death during whole study period (TS)
- Table 3.11.1 Treatment-emergent adverse events leading to discontinuation of study drug during treatment period (TS)
  - Table 3.11.2 Treatment-emergent adverse events leading to discontinuation of study drug during rollover study (TS, patients continuing in the rollover study)
  - Table 3.11.3 Treatment-emergent adverse events leading to discontinuation of study drug during whole study period (TS)
- Table 3.12.1 Treatment-emergent adverse events related to study drug and leading to death during treatment period (TS)
  - Table 3.12.2 Treatment-emergent adverse events related to study drug and leading to death during rollover study (TS, patients continuing in the rollover study)
  - Table 3.12.3 Treatment-emergent adverse events related to study drug and leading to death during whole study period (TS)
  - Table 3.13.1 Non-serious treatment-emergent adverse events occurred at a frequency of  $\geq$ 5% during treatment period (TS)
  - Table 3.13.1 Non-serious treatment-emergent adverse events occurred at a frequency of  $\geq$ 5% during rollover study (TS, patients continuing in the rollover study)
  - Table 3.13.1 Non-serious treatment-emergent adverse events occurred at a frequency of  $\geq$ 5% during whole study period (TS)
  - Table 3.14 Deaths
  - Table 3.15 Urine pregnancy test (TS, women of childbearing potential)
  - Table 3.16 Hematology. Descriptive statistics (TS)
  - Table 3.17 Blood chemistry. Descriptive statistics (TS)
  - Table 3.18 Hematology. Shift table (TS)
  - Table 3.19 Blood chemistry. Shift table (TS)
  - Table 3.20 Hematology. Out of range. Frequency table
  - Table 3.21 Blood chemistry. Out of range. Frequency table (TS)



Table 3.22 Vital signs. Descriptive statistics (TS)

Table 3.23 Vital signs. Out of range. Frequency table (TS)

Table 3.24 Weight. Descriptive statistics (TS)

Table 3.25 ECG. Descriptive statistics (TS)

Table 3.26 ECG. Out of range and General Assessment. Frequency table (TS)

Table 3.27 Physical examinations. Frequency table (TS)



## **Patients Disposition**

F. Hoffmann-La Roche Ltd ML39355

#### Table 1.1 Patients disposition

All Enrolled patients
Page X of X

| | Total |
|---|---|
| | (N = XX) |
| | n (%) |
| Patients who signed the Informed Consent Form | XX |
| Screening Failures | XX |
| Reasons for premature discontinuation | XX |
| Patient request or withdrawal of consent | XX |
| Presence or development of Inclusion/Exclusion criterion (-a) | XX |
| Allocated to treatment | XX |
| Treated during the treatment period | XX (XX.X) |
| Patients continuing (treated) in the rollover study | XX (XX.X) |
| Completed | XX (XX.X) |
| Terminated Prematurely | XX (XX.X) |
| Reasons for premature discontinuation | |
| Pregnancy | XX (XX.X) |
| Unacceptable tolerability and personal safety profile (e.g. adverse events listed in Section 5.1.2 of Protocol, or serious adverse events related to study treatment) | XX (XX.X) |
| Patient request or withdrawal of consent | XX (XX.X) |
| Any medical condition that the investigator or Sponsor determines may jeopardize the patient's safety if he or she continues in the study | XX (XX.X) |
| Investigator or Sponsor determines it is in the best interest of the patient for other reasons | XX (XX.X) |
| Protocol deviation (at Sponsor's discretion) (e.g. refusal to follow study requirements) | XX (XX.X) |
| Termination of the whole study by the Sponsor | XX (XX.X) |
| Lung transplantation | XX (XX.X) |
| The incidence or severity of adverse events in this or other ongoing studies of pirfenidone indicates a potential health hazard to patients | XX (XX.X) |
| Patient enrollment is unsatisfactory | XX (XX.X) |
| Administrative and regulatory reasons | XX (XX.X) |
| Presence or development of Inclusion/Exclusion criterion (-a) | XX (XX.X) |
| Other | XX (XX.X) |

Data extracted: DD.MM.YYYY



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| Other reason 1 | XX (XX.X) |
|----------------|-----------|
| Other reason 2 | XX (XX.X) |
| • • • | XX (XX.X) |

N: the number of patients who signed the Informed Consent Form.

Path to the program code, date and time of output

n: the number of patients within a specific category. Percentages are calculated based on number of patients Allocated to Treatment.



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.2 Violation of eligibility criteria

Screening Failures
Page X of X

| | Total |
|-----------------------------------------------------|----------|
| | (N = XX) |
| | n |
| Patients with any violation of eligibility criteria | XX |
| Patients with any violation of inclusion criteria | XX |
| Inclusion criterion #1 | XX |
| Inclusion criterion #2 | XX |
| ••• | |
| Patients with any violation of exclusion criteria | XX |
| Exclusion criterion #1 | XX |
| Exclusion criterion #2 | XX |
| ••• | ••• |

N: the number of Screening Failures.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

n: the number of patients within a specific category.
Data extracted: DD.MM.YYYY



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Table 1.3 Analysis populations

Allocated to treatment set Page X of X

| | Total |
|--------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Allocated to treatment | XX (100%) |
| Treated set (TS) | XX (XX.X) |
| Full analysis set (FAS) | XX (XX.X) |
| Completed case set (CCS) | XX (XX.X) |

N: the number of patients in the Allocated to treatment set.

n: the number of patients within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

Treated set: patients from 'Allocated to treatment' set, who received any dose of the study treatment.

Full analysis set: patients from 'Treated' set, who had data for at least one post-baseline assessment of any efficacy measurement. Completed case set: patients from 'Full analysis' set, who provided FVC data at 26-week assessment.

Path to the program code, date and time of output



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.4 Study visits

Allocated to treatment set Page X of X

| | Total | Within visit<br>window<br>n (%) |
|---|---|---|
| | (N = XX) | |
| | n (%) | |
| Treatment period | | |
| Start of Treatment (Day 1) | XX (XX.X) | N/A |
| Week 1 Telephone Assessment (+/- 1 day) | XX (XX.X) | XX (XX.X) |
| Week 2 (+/- 2 days) | XX (XX.X) | XX (XX.X) |
| Week 4 (+/- 2 days) | XX (XX.X) | XX (XX.X) |
| Week 8 (+/- 2 days) | XX (XX.X) | XX (XX.X) |
| Week 12 (+/- 2 days) | XX (XX.X) | XX (XX.X) |
| Week 16 (+/- 1 week) | XX (XX.X) | XX (XX.X) |
| Week 20 (+/- 1 week) | XX (XX.X) | XX (XX.X) |
| 1st day at Week 26 (+/- 1 week) | XX (XX.X) | XX (XX.X) |
| 2nd day at Week 26 (+/- 1 week) | XX (XX.X) | XX (XX.X) |
| Follow-up Visit (14-28 days after last dosing) | XX (XX.X) | XX (XX.X) |
| Long Term Follow-Up/Rollover Study | | |
| Week 39 (+/- 2 weeks) | XX (XX.X) | XX (XX.X) |
| Week 52 (+/- 2 weeks) | XX (XX.X) | XX (XX.X) |

N: the number of patients in the Allocated to treatment set.

n: the number of patients within a specific category. Percentages are calculated as (100 x n/N).

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

#### **Protocol Deviations**

F. Hoffmann-La Roche Ltd ML39355

#### Table 1.5 Protocol deviations / violations

Allocated to treatment set
Page X of X

| Total |
|-----------|
| (N = XX) |
| n (%) |
| XX (XX.X) |

N: the number of patients in the Allocated to treatment set.

n: the number of patients with at least one protocol deviation. Percentages are calculated as  $(100 \times n/N)$ .

Path to the program code, date and time of output



## **Demographic and Anthropometric characteristics**

F. Hoffmann-La Roche Ltd ML39355

#### Table 1.6 Demographic characteristics

Treated set Page X of X

| | | Total (N = XX) |
|-------------------|-------|----------------|
| Age, years | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.XX |
| Median | | XX.X |
| Min | | XX |
| Max | | XX |
| Sex | | |
| n | | XX |
| Male | n (%) | XX (XX.X) |
| Female | n (%) | XX (XX.X) |
| Race | | |
| n | | XX |
| Caucasian | n (%) | XX (XX.X) |
| Asian | n (%) | XX (XX.X) |
| Black | n (%) | XX (XX.X) |
| Other | n (%) | XX (XX.X) |
| Other race 1 | n (%) | XX (XX.X) |
| Other race 2 | n (%) | XX (XX.X) |
| ••• | ••• | ••• |
| Ethnicity | | |
| n | | XX |
| Russian | n (%) | XX (XX.X) |
| Tatar | n (%) | XX (XX.X) |
| Ukrainian | n (%) | XX (XX.X) |
| Bashkir | n (%) | XX (XX.X) |
| Chuvash | n (%) | XX (XX.X) |
| Unknown | n (%) | XX (XX.X) |
| Other | n (%) | XX (XX.X) |
| Other ethnicity 1 | n (%) | XX (XX.X) |
| Other ethnicity 2 | n (%) | XX (XX.X) |





N: the number of patients in the Treated set.

n: the number of valid measurements or the number of patients within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

Path to the program code, date and time of output



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.7 Anthropometric characteristics

Treated set Page X of X

| | Total |
|-----------------------------|----------|
| | (N = XX) |
| Height, cm | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min | XX |
| Max | XX |
| Weight, kg | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min | XX |
| Max | XX |
| ody Mass Index (BMI), kg/m2 | XX |
| n | XX.XX |
| Mean | XX.XXX |
| SD | XX.XX |
| Median | XX.X |
| Min | XX.X |
| Max | |

N: the number of patients in the Treated set.

n: the number of valid measurements.

Path to the program code, date and time of output



#### **Baseline Variables**

F. Hoffmann-La Roche Ltd ML39355

#### Table 1.8 Surgical lung biopsy

Treated set Page X of X

| | Total |
|---------------------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Assessment of regional specialist | |
| UIP Pattern | |
| n' | XX |
| Consistent UIP pattern | XX (XX.X) |
| Probable UIP pattern | XX (XX.X) |
| Possible UIP pattern | XX (XX.X) |
| Inconsistent/unclassified UIP pattern | XX (XX.X) |
| Assessment of central specialist | |
| UIP Pattern | |
| n' | XX |
| Consistent UIP pattern | XX (XX.X) |
| Probable UIP pattern | XX (XX.X) |
| Possible UIP pattern | XX (XX.X) |
| Inconsistent/unclassified UIP pattern | XX (XX.X) |

N: the number of patients in the Treated set.  $n^\prime$  - the number of valid observations.

Path to the program code, date and time of output

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.9 HRCT for patient eligibility confirmation

Treated set Page X of X

| | Total |
|-----------------------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Assessment of regional CT-specialist | |
| UIP Pattern | |
| n' | XX |
| Typical (apparent) UIP pattern | XX (XX.X) |
| Possible UIP Pattern | XX (XX.X) |
| Assessment of central CT-specialist (1) | |
| UIP Pattern | |
| n' | XX |
| Typical (apparent) UIP pattern | XX (XX.X) |
| Possible UIP Pattern | XX (XX.X) |
| Inconsistent with UIP Pattern | XX (XX.X) |
| Assessment of central CT-specialist (2) | |
| UIP Pattern | |
| n' | XX |
| Typical (apparent) UIP pattern | XX (XX.X) |
| Possible UIP Pattern | XX (XX.X) |
| Inconsistent with UIP Pattern | XX (XX.X) |
| Not Performed | XX (XX.X) |

N: the number of patients in the Treated set.  $n^{\prime}$  - the number of valid observations.

Path to the program code, date and time of output

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.10 Carbon monoxide diffusing capacity (DLCO)

Treated set Page X of X

| | Total (N = XX) |
|----------------------|----------------|
| Predicted DLCO, % | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min | XX |
| Max | XX |
| Hb-corrected DLCO, % | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min | XX |
| Max | XX |

N: the number of patients in the Treated set.

n: the number of valid measurements.

Path to the program code, date and time of output



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.11 Pre- and post-bronchodilator spirometry parameters at screening

Treated set Page X of X

| | Total |
|------------------------------|----------|
| | (N = XX) |
| Pre-bronchodilator FEV1/FVC | |
| n | XX |
| Mean | XX.XX |
| SD | XX.XXX |
| Median | XX.XX |
| Min | XX.XX |
| Max | XX.XX |
| Post-bronchodilator FEV1/FVC | |
| n | XX |
| Mean | XX.XX |
| SD | XX.XXX |
| Median | XX.XX |
| Min | XX.XX |
| Max | XX.XX |
| ••• | |

N: the number of patients in the Treated set.

n: the number of valid measurements.

Path to the program code, date and time of output

<Table will be continued for Pre-, post- bronchodilator FVC (absolute), ml; FVC (relative), % predicted>



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.12 Serologic tests

Treated set Page X of X

| | Total |
|----------------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Rheumatoid factor | |
| n' | XX |
| Positive | XX (XX.X) |
| Negative | XX (XX.X) |
| Anticyclic citrullinated peptide | |
| n' | XX |
| Positive | XX (XX.X) |
| Negative (<= 5 U/ml) | XX (XX.X) |
| Antinuclear antibody titer | |
| n' | XX |
| Positive | XX (XX.X) |
| Negative | XX (XX.X) |

N: the number of patients in the Treated set. n': the number of valid observations.

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.

Path to the program code, date and time of output



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.13 GAP assessment

Treated set Page X of X

| | | Total $(N = XX)$ |
|------------------------------|-------|------------------|
| GAP index | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.XX |
| Median | | XX.X |
| Min | | XX |
| Max | | XX |
| Stage | | |
| n <b>'</b> | | XX |
| I | n (%) | XX (XX.X) |
| II | n (%) | XX (XX.X) |
| III | n (%) | XX (XX.X) |
| Individual risk of mortality | | |
| One year (1-yr) mortality | | |
| n | | XX |
| Mean | | XX.XX |
| SD | | XX.XXX |
| Median | | XX.XX |
| Min | | XX.X |
| Max | | XX.X |
| Two year (2-yr) mortality | | |
| n | | XX |
| Mean | | XX.XX |
| SD | | XX.XXX |
| Median | | XX.XX |
| Min | | XX.X |
| Max | | XX.X |
| Three year (3-yr) mortality | | |
| n | | XX |
| Mean | | XX.XX |

Data extracted: DD.MM.YYYY



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| SD | XX.XXX |
|--------|--------|
| Median | XX.XX |
| Min | XX.X |
| Max | XX.X |

N: the number of patients in the Treated set. n': the number of valid observations.

Path to the program code, date and time of output

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.14 Review transbronchial lung biopsy/BAL

Treated set Page X of X

| | Total (N = XX) |
|---|---|
| | n (%) |
| Are there features supporting an alternative diagnosis after review transbronchial lung biopsy? | |
| n' | XX |
| Yes | XX (XX.X) |
| No | XX (XX.X) |
| Are there features supporting an alternative diagnosis after review BAL? | XX (XX.X) |
| n' | XX |
| Yes | XX (XX.X) |
| No | XX (XX.X) |

N: the number of patients in the Treated set.  ${\rm n}^\prime$  - the number of valid observations.

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.

Path to the program code, date and time of output



#### **Medical history**

F. Hoffmann-La Roche Ltd ML39355

#### Table 1.15 Prior medical/surgical conditions/diagnoses

Treated set Page X of X

| System Organ Class (SOC) | Total |
|--------------------------|-----------------------|
| Preferred Term (PT) | (N = XX)<br>n (%) / E |
| Overall | xx (xx.x) / xx |
| System Organ Class 1 | XX (XX.X) / XX |
| Preferred Term 1 | XX (XX.X) / XX |
| Preferred Term 2 | XX (XX.X) / XX |
| | ••• |
| ystem Organ Class 2 | XX (XX.X) / XX |
| Preferred Term 1 | XX (XX.X) / XX |
| Preferred Term 2 | XX (XX.X) / XX |
| ••• | ••• |
| •• | ••• |

N: the number of patients in the Treated set.

Medical history events are coded using MedDRA version XX.X.

Each patient is counted only once per preferred term (PT) and once per system organ class (SOC).

Path to the program code, date and time of output

<System organ classes (SOC) and preferred terms (PT) within each SOC are sorted in descending order of n(%).>

n: the number of patients with at least one  $\underline{\text{prior}}$  medical history event within a specific category. Percentages are calculated as (100 x n/N).

E: total number of prior medical history events reported within a specific category.



Similar to table 1.15, the following tables will be constructed (with corrections of underlined fragments in the note):

F. Hoffmann-La Roche Ltd ML39355

Table 1.16 Concurrent medical/surgical conditions/diagnoses

Treated set Page X of X



F. Hoffmann-La Roche Ltd ML39355

#### Table 1.17 History of idiopathic pulmonary fibrosis

Treated set Page X of X

| | | Total |
|---|---|---|
| | | (N = XX) |
| Duration of clinical symptoms consistent with IPF, months | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.XX |
| Median | | XX.X |
| Min | | XX |
| Max | | XX |
| Clinically significant environmental exposure known to cause | pulmonary fibrosis | |
| n' | 1 | XX |
| Yes | n (%) | XX (XX.X) |
| No | n (%) | XX (XX.X) |
| Known explanation for interstitial lung disease | | |
| n' | | XX |
| Yes | n (%) | XX (XX.X) |
| No | n (%) | XX (XX.X) |
| Cigarette smoking within 28 days before the treatment start | | |
| n' | | XX |
| Yes | n (%) | XX (XX.X) |
| No | n (%) | XX (XX.X) |

N: the number of patients in the Treated set.

Path to the program code, date and time of output

n: the number of patients within a specific category.  $n^{\prime}$  - the number of valid observations.

Percentages are based on the corresponding number of valid observations.



#### Prior and concomitant medications

F. Hoffmann-La Roche Ltd ML39355

#### Table 1.18 Prior medications

Treated set Page X of X

| Pharmacological subgroup (3rd level) Chemical substance (5th level) | Total<br>(N = XX)<br>n (%) / E |
|---|---|
| Overall | XX (XX.X) / XX |
| Pharmacological subgroup 1 Chemical substance 1 Chemical substance 2 | XX (XX.X) / XX<br>XX (XX.X) / XX<br>XX (XX.X) / XX |
| Pharmacological subgroup 2 Chemical substance 1 Chemical substance 2 | XX (XX.X) / XX<br>XX (XX.X) / XX<br>XX (XX.X) / XX |
| | ••• |

N: the number of patients in the Treated set.

Medications are coded by WHO drug dictionary version XX.X.

Path to the program code, date and time of output

<The pharmacological subgroups and chemical substances within each pharmacological subgroup are sorted in descending order of n (%). Each patient is
counted only once per pharmacological subgroup and once per chemical substance.>

n: the number of patients with at least one prior medication within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

E: total number of prior medications reported within a specific category.



Similar to table 1.18, the following tables will be constructed (with corrections of underlined fragments in the note):

F. Hoffmann-La Roche Ltd ML39355

Table 1.19 Concomitant medications

Treated set Page X of X

F. Hoffmann-La Roche Ltd ML39355

Table 1.20 Concomitant medications during rollover study Treated set (patients continuing in the rollover study) Page X of X



## **Efficacy Analyses**

#### **Primary Efficacy Endpoint**

# F. Hoffmann-La Roche Ltd ML39355

#### Table 2.1 Descriptive statistics for FVC by visit

Full analysis set (FAS)
Page X of X

Parameter: XXXXXXXXX, <units>

| | Total (N = XX) | Change from the baseline |
|---------------|--------------------|--------------------------|
| Screening | | |
| n | XX | |
| Mean [95% CI] | xx.x [xx.x - xx.x] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Day 1 | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Baseline | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 12 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X = XX.X = XX.X | XX.X [XX.X - XX.X] |



| SD | XX.XX | XX.XX |
|---------------|--------------------|--------------------|
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 12* | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 52 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 52* | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |

N: the number of patients in the FAS.

Baseline FVC is the average of the pre-bronchodilator FVC measured at the Screening and Day 1 visits. The FVC at Week 26 is the average of the FVC measured on two separate days at Week 26.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

<Report the following assessments: Screening (pre-bronchodilator), Day 1, Baseline, Week 12, Week 26 Day 1, Week 26 Day 2, Week 39, Week 52> <FVC values within the visit window will also be presented descriptively for the following assessments: Week 12\*, Week 26 Day 1\*, Week 26 Day 2\*, Week 26\*, Week 39\*, Week 52\*>

<Report the following parameters: FVC (absolute), mL/ FVC (relative) predicted, %>

n: the number of valid measurements.

<sup>\*:</sup> Values assessed within the corresponding visit window.



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.2 Primary efficacy endpoint

Full analysis set (FAS)
Page X of X

Parameter: XXXXXXXXX, <units>

| | Total (N = XX) | Change from the baseline |
|---|---|---|
| Baseline | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 26, Primary analysis | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 26, Sensitivity analysis 1 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 26, Sensitivity analysis 2 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |

N: the number of patients in the FAS.

Data extracted: DD.MM.YYYY



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

n: the number of valid measurements.

Baseline FVC is the average of the pre-bronchodilator FVC measured at the Screening and Day 1 visits. The FVC at Week 26 is the average of the FVC measured on two separate days at Week 26.

Sensitivity analyses 1 - 6 related to missing Week 26 data imputation are described in SAP Section 8.1; Sensitivity analysis 7 - Primary analysis excluding all FVC values outside of visit window. Sensitivity analysis 8 - Complete case set; Sensitivity analysis 9 - Complete case set excluding all FVC values outside of visit window.

Path to the program code, date and time of output

<Report the following parameters: FVC (absolute), mL/ FVC (relative) predicted, %>



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.3 Primary efficacy endpoint: categorical results

Full analysis set (FAS)
Page X of X

Parameter: XXXXXXXXX, <units> <[1]/[2]>

| | Total $(N = XX)$ |
|---|---|
| | n (%) |
| Week 26, Primary analysis | |
| n' | XX |
| Patients with decline of $\geq$ 10% from Baseline or death before Week 26 | XX (XX.X) |
| Decline of < 10% to 0% | XX (XX.X) |
| Patients with improvement of ≥0% from Baseline | XX (XX.X) |
| Week 26, Sensitivity analysis 1 | |
| n' | XX |
| Patients with decline of $\geq$ 10% from Baseline or death before Week 26 | XX (XX.X) |
| Decline of < 10% to 0% | XX (XX.X) |
| Patients with improvement of ≥0% from Baseline | XX (XX.X) |
| Week 26, Sensitivity analysis 2 | |
| n' | XX |
| Patients with decline of $\geq$ 10% from Baseline or death before Week 26 | XX (XX.X) |
| Decline of < 10% to 0% | XX (XX.X) |
| Patients with improvement of $\geq$ 0% from Baseline | XX (XX.X) |

N: the number of patients in the FAS. n: the number of patients within a specific category. n': the number of valid observations. Percentages are based on the corresponding number of valid observations.

[1] Percentage change (Week 26 FVC value - Baseline FVC)\*100/ Baseline FVC; [2] Absolute change in FVC % predicted.

Baseline FVC is the average of the pre-bronchodilator FVC measured at the Screening and Day 1 visits. The FVC at Week 26 is the average of the FVC measured on two separate days at Week 26.

Sensitivity analyses 1 - 6 related to missing Week 26 data imputation are described in SAP Section 8.1; Sensitivity analysis 7 - Primary analysis excluding all FVC values outside of visit window. Sensitivity analysis 8 - Complete case set; Sensitivity analysis 9 - Complete case set excluding all FVC values outside of visit window.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

<Report the following parameters: FVC (absolute), mL [1]/ FVC (relative) predicted, % [2]>



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.4 Primary efficacy endpoint by pattern type

Complete case set (CCS)
Page X of X

Parameter: XXXXXXXXX, <units>

| | Total (N = XX) | Change from the baseline |
|--------------------|--------------------|--------------------------|
| Baseline | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Baseline Pattern 1 | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Baseline Pattern 2 | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 26 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 26, Pattern 1 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |

Data extracted: DD.MM.YYYY



#### ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| SD | XX.XX | XX.XX |
|--------------------|--------------------|--------------------|
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 26, Pattern 2 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |

 ${\tt N:}$  the number of patients in the CCS.  ${\tt n:}$  the number of valid measurements.

Baseline FVC is the average of the pre-bronchodilator FVC measured at the Screening and Day 1 visits. The FVC at Week 26 is the average of the FVC measured on two separate days at Week 26.

Pattern 1: Patients who received study drug until 26 weeks;

Pattern 2: Patients who prematurely discontinued study drug, but who were followed up until Week 26.

Path to the program code, date and time of output



## **Secondary Efficacy Endpoint**

#### **6-Minute Walk Test**

F. Hoffmann-La Roche Ltd ML39355

#### Table 2.5 6-Minute Walk Test

Full analysis set (FAS)
Page X of X

| | Total $(N = XX)$ | Change from the baseline |
|-----------------------|--------------------|--------------------------|
| 6-Minute Walk Test, m | | |
| Screening | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Day 1 | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Baseline | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 12 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |



| Max | XX | XX |
|---------------|--------------------|--------------------|
| Week 12* | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Week 52 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX .XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 52* | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |

N: the number of patients in the FAS.

Baseline 6MWT distance is the average of the measurements measured at the Screening and Day 1 visits. The 6MWT distance at Week 26 is defined as the average of the 6MWT distance measured on two separate days at Week 26.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

<The following assessments will be presented: Screening, Day 1, Baseline, Week 12, Week 26 Day 1, Week 26 Day 2, Week 26, Week 39, Week 52>
<Values within the visit window will also be presented descriptively for the following assessments: Week 12\*, Week 26 Day 1\*, Week 26 Day 2\*, Week 26\*,
Week 39\*, Week 52\*>

n: the number of valid measurements.

<sup>\*:</sup> Values assessed within the corresponding visit window.



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.6 Change in 6MWT distance at Week 26 by category

Full analysis set (FAS)
Page X of X

| | Total |
|---|---|
| | (N = XX) |
| | n (%) |
| n' | XX |
| Patients with decline of $\geq$ 50 m from Baseline or death before Week 26 | XX (XX.X) |
| Patients with decline of $<$ 50 m to 0 m from Baseline | XX (XX.X) |
| Patients with improvement of ≥0 m from Baseline | XX (XX.X) |

N: the number of patients in the Full analysis set (FAS).  $n^\prime$  - the number of valid observations.

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.

Path to the program code, date and time of output



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.7 Borg scale

Full analysis set (FAS)
Page X of X

| • | $ \begin{array}{ccc} {\tt Total} \\ ({\tt N} = {\tt XX}) \end{array} $ | Change Pre-test from<br>Baseline Pre-test | Change Post-test from<br>Pre-test |
|---|---|---|---|
| Borg scale | | | |
| Screening Pre-test | | | |
| n | XX | | |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | | |
| SD | XX.XXX | | |
| Median | XX.XX | | |
| Min | XX.X | | |
| Max | XX.X | | |
| Screening Post-test | | | |
| n | XX | | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | | XX.XX [XX.XX - XX.XX] |
| SD | XX.XXX | | XX.XXX |
| Median | XX.XX | | XX.XX |
| Min | XX.X | | XX.X |
| Max | XX.X | | XX.X |
| Day 1 Pre-test | | | |
| n | XX | | |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | | |
| SD | XX.XXX | | |
| Median | XX.XX | | |
| Min | XX.X | | |
| Max | XX.X | | |
| Day 1 Post-test | | | |
| n | XX | | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | | XX.XX [XX.XX - XX.XX] |
| SD | XX.XXX | | XX.XXX |
| Median | XX.XX | | XX.XX |
| Min | XX.X | | XX.X |
| Max | XX.X | | XX.X |
| ••• | | | |
| ••• | | | |



| Week 26 Day 1 Pre-test n Mean [95% CI] SD Median Min Max | XX<br>XX.XX [XX.XX - XX.XX]<br>XX.XXX<br>XX.XX<br>XX.X<br>XX.X | xx<br>xx.xx [xx.xx - xx.xx]<br>xx.xxx<br>xx.xx<br>xx.x<br>xx.x<br>xx.x | |
|---|---|---|---|
| Week 26 Day 1 Post-test<br>n<br>Mean [95% CI]<br>SD<br>Median<br>Min<br>Max | XX<br>XX.XX [XX.XX - XX.XX]<br>XX.XXX<br>XX.XX<br>XX.X<br>XX.X | | XX<br>XX.XX [XX.XX - XX.XX]<br>XX.XXX<br>XX.XX<br>XX.X<br>XX.X |
| Week 26* Day 1 Pre-test | XX<br>XX.XX [XX.XX - XX.XX] | XX<br>XX.XX [XX.XX - XX.XX] | |
| Mean [95% CI] SD Median Min | XX.XXX<br>XX.XX<br>XX.X | XX.XXX<br>XX.XX<br>XX.X | |
| Max Week 26* Day 1 Post-test n Mean [95% CI] SD | XX.X XX XX.XX [XX.XX - XX.XX] XX.XXX | XX.X | XX<br>XX.XX [XX.XX - XX.XX]<br>XX.XXX |
| Median<br>Min<br>Max | XX.XX<br>XX.X<br>XX.X | | XX.XX<br>XX.X<br>XX.X |
| Week 52* Post-test n Mean [95% CI] SD Median | <br>XX<br>XX.XX [XX.XX - XX.XX]<br>XX.XXX<br>XX.XX | ••• | <br>xx<br>xx.xx [xx.xx - xx.xx]<br>xx.xxx<br>xx.xx |

Data extracted: DD.MM.YYYY



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| Min | XX.X | XX.X |
|-----|------|------|
| Max | XX.X | XX.X |

N: the number of patients in the FAS.

Baseline Borg scale result is the average of the measurements at the Screening and Day 1 visits. The Borg scale at Week 26 is defined as the average of the Borg scale results measured on two separate days at Week 26.

Path to the program code, date and time of output

<The following assessments will be presented: Screening, Day 1, Baseline, Week 12, Week 26 Day 1, Week 26 Day 2, Week 26, Week 39, Week 52>
<Values within the visit window will also be presented descriptively for the following assessments: Week 12\*, Week 26 Day 1\*, Week 26 Day 2\*, Week 26\*, Week 39\*, Week 52\*>

n: the number of valid measurements.

<sup>\*:</sup> Values assessed within the corresponding visit window.

Total



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

EQ-5D-5L

F. Hoffmann-La Roche Ltd ML39355

#### Table 2.8 EQ-5D-5L. Descriptive statistics

Full analysis set (FAS)
Page X of X

Dimension: <Mobility/ Self-Care/ Usual Activities /Pain/Discomfort/ Anxiety/Depression>

| | Total |
|--------------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Baseline n' | W |
| | XX |
| Level 1 (no problem) | XX (XX.X) |
| Level 2 (slight problems) | XX (XX.X) |
| Level 3 (moderate problems) | XX (XX.X) |
| Level 4 (severe problems) | XX (XX.X) |
| Level 5 (unable to walk about) | XX (XX.X) |
| Week 12 | |
| n' | XX |
| Level 1 (no problem) | XX (XX.X) |
| Level 2 (slight problems) | XX (XX.X) |
| Level 3 (moderate problems) | XX (XX.X) |
| Level 4 (severe problems) | XX (XX.X) |
| Level 5 (unable to walk about) | XX (XX.X) |
| Week 12* | |
| n' | XX |
| Level 1 (no problem) | XX (XX.X) |
| Level 2 (slight problems) | XX (XX.X) |
| Level 3 (moderate problems) | XX (XX.X) |
| Level 4 (severe problems) | XX (XX.X) |
| Level 5 (unable to walk about) | XX (XX.X) |
| Mark 00 | |
| Week 26 n' | XX |
| Level 1 (no problem) | XX (XX.X) |
| Level 2 (slight problems) | XX (XX.X) |
| Level 3 (moderate problems) | XX (XX.X) |
| Level 4 (severe problems) | XX (XX.X) |
| Level 5 (unable to walk about) | XX (XX.X) |
| • • • | |

Data extracted: DD.MM.YYYY



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

N: the number of patients in the Full analysis set (FAS).  $n^\prime$  - the number of valid observations.

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations. Baseline is the last non-missing assessment prior to the first dose of the study drug.

\*: Values assessed within the corresponding visit window.

Path to the program code, date and time of output



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.9 Change in EQ-5D-5L. Mobility

Full analysis set (FAS)
Page X of X

Dimension: <Mobility/ Self-Care/ Usual Activities /Pain/Discomfort/ Anxiety/Depression>

| | Baseline assessment | | | | | |
|---|---|---|---|---|---|---|
| | Level 1 (no problem) n (%) | Level 2 (slight problems) n (%) | Level 3 (moderate problems) n (%) | Level 4 (severe problems) n (%) | Level 5 (unable to<br>walk about)<br>n (%) | Total<br>(N = XX)<br>n (%) |
| Baseline | ( + / | ( * / | ( ) | ( • / | (*) | ( • / |
| Level 1 (no problem) | | | | | | XX (XX.X) |
| Level 2 (slight problems) | | | | | | XX (XX.X) |
| Level 3 (moderate problems) | | | | | | XX (XX.X) |
| Level 4 (severe problems) | | | | | | XX (XX.X) |
| Level 5 (unable to walk about) | | | | | | XX (XX.X) |
| Total | | | | | | XX (100) |
| Week 12 | | | | | | |
| Level 1 (no problem) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 2 (slight problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 3 (moderate problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 4 (severe problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 5 (unable to walk about) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Week 12* | | | | | | |
| • • • | • • • | ••• | • • • | ••• | • • • | • • • |
| Week 52* | | | | | | |
| • • • | | | | | | |

N: the number of patients in the Full analysis set (FAS).

Path to the program code, date and time of output

n: the number of patients within a specific category. Percentages are based on the number of non-missing values at baseline and at the corresponding visit.

Baseline is the last non-missing assessment prior to the first dose of the study drug.

<sup>\*:</sup> Values assessed within the corresponding visit window.



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.10 Change in EQ-5D-5L. Self-Care

Full analysis set (FAS)
Page X of X

Dimension: <Mobility/ Self-Care/ Usual Activities /Pain/Discomfort/ Anxiety/Depression>

| | Baseline assessment | | | | | |
|---|---|---|---|---|---|---|
| | Level 1 (no problem) | m) (slight problems) | Level 3 (moderate problems) | Level 4 (severe problems) n (%) | Level 5 (unable<br>to wash or<br>dress myself)<br>n (%) | Total<br>(N = XX)<br>n (%) |
| | n (%) | | | | | |
| Baseline | | | | | | |
| Level 1 (no problem) | | | | | | XX (XX.X) |
| Level 2 (slight problems) | | | | | | XX (XX.X) |
| Level 3 (moderate problems) | | | | | | XX (XX.X) |
| Level 4 (severe problems) | | | | | | XX (XX.X) |
| Level 5 (unable to wash or dress myself) | | | | | | XX (XX.X) |
| Total | | | | | | XX (100) |
| Week 12 | | | | | | |
| Level 1 (no problem) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 2 (slight problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 3 (moderate problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 4 (severe problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 5 (unable to wash or dress myself) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Week 12* | | | | | | |
| ••• | • • • | • • • | • • • | • • • | • • • | • • • |
| Week 52* | | | | | | |
| • • • | | | | | | |

N: the number of patients in the Full analysis set (FAS).

Path to the program code, date and time of output

F. Hoffmann-La Roche Ltd

n: the number of patients within a specific category. Percentages are based on the number of non-missing values at baseline and at the corresponding visit.

Baseline is the last non-missing assessment prior to the first dose of the study drug.

<sup>\*:</sup> Values assessed within the corresponding visit window.


ML39355

#### Table 2.11 Change in EQ-5D-5L. Usual Activities

Full analysis set (FAS)
Page X of X

Dimension: <Mobility/ Self-Care/ Usual Activities /Pain/Discomfort/ Anxiety/Depression>

| | Baseline assessment | | | | | |
|---|---|---|---|---|---|---|
| | Level 1 (no problem) | Level 2<br>(slight<br>problems) | Level 3 (moderate problems) | Level 4 (severe problems) | Level 5 (unable<br>to do my usual<br>activities) | Total (N = XX) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline | | | | | | |
| Level 1 (no problem) | | | | | | XX (XX.X) |
| Level 2 (slight problems) | | | | | | XX (XX.X) |
| Level 3 (moderate problems) | | | | | | XX (XX.X) |
| Level 4 (severe problems) | | | | | | XX (XX.X) |
| Level 5 (unable to do my usual activities) | | | | | | XX (XX.X) |
| Total | | | | | | XX (100) |
| Week 12 | | | | | | |
| Level 1 (no problem) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 2 (slight problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| Level 3 (moderate problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| Level 4 (severe problems) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| Level 5 (unable to do my usual activities) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Week 12* | | | | | | |
| ••• | • • • | • • • | • • • | ••• | ••• | • • • |
| Week 52* | | | | | | |
| • • • | | | | | | |

N: the number of patients in the Full analysis set (FAS).

Path to the program code, date and time of output

n: the number of patients within a specific category. Percentages are based on the number of non-missing values at baseline and at the corresponding visit.

Baseline is the last non-missing assessment prior to the first dose of the study drug.

<sup>\*:</sup> Values assessed within the corresponding visit window.



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.12 Change in EQ-5D-5L. Pain/Discomfort

Full analysis set (FAS)
Page X of X

Dimension: <Mobility/ Self-Care/ Usual Activities /Pain/Discomfort/ Anxiety/Depression>

| | Baseline assessment | | | | | |
|---|---|---|---|---|---|---|
| | Level 1 (no pain or discomfort) n (%) | Level 2 (slight pain or discomfort) n (%) | Level 3 (moderate pain or discomfort) n (%) | Level 4 (severe pain or discomfort) n (%) | Level 5 (extreme pain or discomfort) n (%) | Total (N = XX) n (%) |
| Baseline | | | | | | |
| Level 1 (no pain or discomfort) | | | | | | XX (XX. |
| Level 2 (slight pain or discomfort) | | | | | | XX (XX. |
| Level 3 (moderate pain or discomfort) | | | | | | XX (XX. |
| Level 4 (severe pain or discomfort) | | | | | | XX (XX. |
| Level 5 (extreme pain or discomfort) | | | | | | XX (XX. |
| Total | | | | | | XX (100 |
| Week 12 | | | | | | |
| Level 1 (no pain or discomfort) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX. |
| Level 2 (slight pain or discomfort) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX. |
| Level 3 (moderate pain or discomfort) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX. |
| Level 4 (severe pain or discomfort) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX. |
| Level 5 (extreme pain or discomfort) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX. |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100 |
| Week 12* | | | | | | |
| ••• | • • • | • • • | • • • | • • • | • • • | |
| Week 52* | | | | | | |
| • • • | | | | | | |

N: the number of patients in the Full analysis set (FAS).

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

F. Hoffmann-La Roche Ltd

n: the number of patients within a specific category. Percentages are based on the number of non-missing values at baseline and at the corresponding visit.

Baseline is the last non-missing assessment prior to the first dose of the study drug.

<sup>\*:</sup> Values assessed within the corresponding visit window.



ML39355

#### Table 2.13 Change in EQ-5D-5L. Anxiety/Depression

Full analysis set (FAS)
Page X of X

Dimension: <Mobility/ Self-Care/ Usual Activities /Pain/Discomfort/ Anxiety/Depression>

| | Baseline assessment | | | | | |
|---|---|---|---|---|---|---|
| | Level 1 (not anxious or depressed) | Level 2 (slight anxious or depressed) | Level 3 (moderate anxious or depressed) | Level 4 (severe anxious or depressed) | Level 5 (extremely anxious or depressed) | Total (N = XX) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline | | | | | | |
| Level 1 (not anxious or depressed) | | | | | | XX (XX.X) |
| Level 2 (slight anxious or depressed) | | | | | | XX (XX.X) |
| Level 3 (moderate anxious or depressed) | | | | | | XX (XX.X) |
| Level 4 (severe anxious or depressed) | | | | | | XX (XX.X) |
| Level 5 (extremely anxious or depressed) | | | | | | XX (XX.X) |
| Total | | | | | | XX (100) |
| Week 12 | | | | | | |
| Level 1 (not anxious or depressed) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 2 (slight anxious or depressed) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 3 (moderate anxious or depressed) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 4 (severe anxious or depressed) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Level 5 (extremely anxious or depressed) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Week 12* | | | | | | |
| ••• | • • • | • • • | ••• | • • • | • • • | • • • |
| Week 52* | | | | | | |
| ••• | | | | | | |

N: the number of patients in the Full analysis set (FAS).

Path to the program code, date and time of output

n: the number of patients within a specific category. Percentages are based on the number of non-missing values at baseline and at the corresponding visit.

Baseline is the last non-missing assessment prior to the first dose of the study drug.

<sup>\*:</sup> Values assessed within the corresponding visit window.



F. Hoffmann-La Roche Ltd ML39355

### Table 2.14 EQ-5D-5L. VAS and Index score

Full analysis set (FAS)
Page X of X

Parameter: XXXXXXXXX

| arameter. AAAAAAAA | Total $(N = XX)$ | Change from the baseline |
|--------------------|------------------|--------------------------|
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 12* | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| ••• | | |
| Week 52* | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |





N: the number of patients in the FAS.

n: the number of valid measurements.

Baseline is the last non-missing assessment prior to the first dose of the study drug.

\*: Values assessed within the corresponding visit window.

Path to the program code, date and time of output



## **Exploratory Efficacy Endpoint**

F. Hoffmann-La Roche Ltd ML39355

### Table 2.15 HRCT. HRCT fibrosis score

Full analysis set (FAS)
Page X of X

| | Total (N = XX) | Change from the baseline |
|---|---|---|
| HRCT fibrosis score | | |
| Baseline | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 26 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 52 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| p-value for (Week 26 - Baseline) comparison | 0.XXXX | |
| p-value for (Week 52 - Baseline) comparison | 0.XXXX | |

N: the number of patients in the FAS.

n: the number of valid measurements.

The comparison of the results is performed using the paired t-test.





Path to the program code, date and time of output

Data extracted: DD.MM.YYYY



F. Hoffmann-La Roche Ltd ML39355

### Table 2.16 HRCT. Lung opacity score

Full analysis set (FAS)
Page X of X

| | Total $(N = XX)$ | Change from the baseline |
|--------------------|--------------------|--------------------------|
| Lung opacity score | | |
| Baseline | | |
| n | XX | |
| Mean [95% CI] | XX.X [XX.X - XX.X] | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 26 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| Week 52 | | |
| n | XX | XX |
| Mean [95% CI] | XX.X [XX.X - XX.X] | XX.X [XX.X - XX.X] |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |

N: the number of patients in the FAS.

Path to the program code, date and time of output

n: the number of valid measurements.



F. Hoffmann-La Roche Ltd ML39355

#### Table 2.17 Exacerbation cases during treatment period

Full analysis set (FAS)
Page X of X

| System Organ Class (SOC) Preferred Term (PT) | Total<br>(N = XX)<br>n (%) / E |
|---|---|
| Overall | XX (XX.X) / XX |
| System Organ Class 1 | XX (XX.X) / XX |
| Preferred Term 1 | XX (XX.X) / XX |
| Preferred Term 2 | XX (XX.X) / XX |
| • • • | |
| System Organ Class 2 | XX (XX.X) / XX |
| Preferred Term 1 | XX (XX.X) / XX |
| Preferred Term 2 | XX (XX.X) / XX |
| ••• | ••• |

N: the number of patients in the FAS. E: number of adverse events reported.

n: the number of patients within the corresponding category. Percentages are calculated as  $100 \times (n/N)$ .

Adverse events were coded using the MedDRA version XX.X.

Each patient is counted only once per preferred term (PT) and once per system organ class (SOC).

<System organ classes (SOC) and preferred terms (PT) within each SOC should be sorted in descending order of n(%).>

Path to the program code, date and time of output



Similar to table 2.17, the following tables will be constructed:

F. Hoffmann-La Roche Ltd ML39355

### Table 2.18 Exacerbation cases during rollover study

Full analysis set (FAS, patients continuing in the rollover study)  $\hspace{1.5cm} \text{Page X of X}$ 

F. Hoffmann-La Roche Ltd ML39355

### Table 2.19 Exacerbation cases during whole study period

Full analysis set (FAS, patients continuing in the rollover study) Page X of X



### **Safety Analyses**

## **Exposure**

F. Hoffmann-La Roche Ltd ML39355

### Table 3.1 Duration of exposure

Treated set (TS)
Page X of X

| | | Total (N = XX) |
|---|---|---|
| Duration of exposure to Pirfenidone dur | ing treatment period, weeks | (14 2727) |
| n | | XX |
| Mean | | XX.XX |
| SD | | XX.XXX |
| Median | | XX.XX |
| Min | | XX.X |
| Max | | XX.X |
| Duration of exposure to Pirfenidone dur | ing rollover study, weeks | |
| n | | XX |
| Mean | | XX.XX |
| SD | | XX.XXX |
| Median | | XX.XX |
| Min | | XX.X |
| Max | | XX.X |
| Total duration of exposure to Pirfenio | done (only for patients continuing in the rollover study), weeks | |
| | | XX |
| n | | $\Delta\Delta$ |
| n<br>Mean | | |
| Mean | | XX.XX |
| Mean<br>SD | | |
| Mean | | XX.XX<br>XX.XXX |

N: the number of patients in the Treated set (TS).

n: the number of valid measurements.





Path to the program code, date and time of output

Data extracted: DD.MM.YYYY



F. Hoffmann-La Roche Ltd ML39355

### Table 3.2 Total number of capsules taken

Treated set (TS)
Page X of X

| | Total (N = XX) |
|---|---|
| Total number of capsules taken during treatment period | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min | XX |
| Max | XX |
| Total number of capsules taken during rollover study | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min | XX |
| Marr | |
| Max | XX |
| Total number of capsules taken during the study (only for page 1) | |
| Total number of capsules taken during the study (only for pa | atients continuing in the rollover study) |
| Total number of capsules taken during the study (only for particles of the study o | atients continuing in the rollover study) XX |
| Total number of capsules taken during the study (only for page of the study) notes that the study of the stud | atients continuing in the rollover study) XX XX.X |
| Total number of capsules taken during the study (only for page of the study) of the study (only for page of the st | atients continuing in the rollover study) XX XX.X XX.XX |

N: the number of patients in the Treated set (TS).

Path to the program code, date and time of output

n: the number of valid measurements.





### **Adverse Events**

F. Hoffmann-La Roche Ltd ML39355

### Table 3.3.1 Treatment-emergent adverse events during treatment period

Treated set (TS) Page X of X

| System Organ Class (SOC) Preferred Term (PT) | Total<br>(N = XX)<br>n (%) / E |
|---|---|
| Overall | XX (XX.X) / XX |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | XX (XX.X) / XX<br>XX (XX.X) / XX<br>XX (XX.X) / XX |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | XX (XX.X) / XX<br>XX (XX.X) / XX<br>XX (XX.X) / XX |

N: the number of patients in the Treated set (TS).

Each patient is counted only once per preferred term (PT) and once per system organ class (SOC).

Adverse events are coded by MedDRA version XX.X.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

<System organ classes (SOC) and preferred terms (PT) within each SOC should be sorted in descending order of n (%). >

n: the number of patients with at least one TEAE within a specific category. Percentages are calculated as (100 x n/N).

E: total number of TEAEs reported within a specific category.



Similar to table 3.3.1, the following tables will be constructed (with the corresponding corrections of underlined fragments in the note):

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.3.2 Treatment-emergent adverse events during rollover study

Treated set (TS, patients continuing in the rollover study)  $Page \ X \ of \ X$ 

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.3.3 Treatment-emergent adverse events during whole study period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd ML39355

### Table 3.4.1 Treatment-emergent adverse events related to the study drug during treatment period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.4.2 Treatment-emergent adverse events related to the study drug during rollover study

> F. Hoffmann-La Roche Ltd ML39355

#### Table 3.4.3 Treatment-emergent adverse events related to the study drug during whole study period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.5.1 Serious treatment-emergent adverse events during treatment period

Treated set (TS)
Page X of X



F. Hoffmann-La Roche Ltd ML39355

Table 3.5.2 Serious treatment-emergent adverse events during rollover study

Treated set (TS, patients continuing in the rollover study) Page X of X

F. Hoffmann-La Roche Ltd ML39355

Table 3.5.3 Serious treatment-emergent adverse events during whole study period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd ML39355

Table 3.6.1 Serious treatment-emergent adverse events related to the study drug during treatment period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.6.2 Serious treatment-emergent adverse events related to the study drug during rollover study

F. Hoffmann-La Roche Ltd

ML39355

Table 3.6.3 Serious treatment-emergent adverse events related to the study drug during whole study period

Treated set (TS)
Page X of X



F. Hoffmann-La Roche Ltd ML39355

Table 3.7.1 Treatment-emergent adverse events during treatment period by maximum severity Treated set (TS)

Page X of X

| System Organ Class (SOC) | | Total |
|--------------------------|----------|----------------|
| Preferred Term (PT) | Severity | (N = XX) |
| Fieleffed Term (F1) | | n (%) / E |
| Overall | Grade 1 | XX (XX.X) / XX |
| | Grade 2 | XX (XX.X) / XX |
| | Grade 3 | XX (XX.X) / XX |
| | Grade 4 | XX (XX.X) / XX |
| | Grade 5 | XX (XX.X) / XX |
| System Organ Class 1 | Grade 1 | XX (XX.X) / XX |
| | Grade 2 | XX (XX.X) / XX |
| | Grade 3 | XX (XX.X) / XX |
| | Grade 4 | XX (XX.X) / XX |
| | Grade 5 | XX (XX.X) / XX |
| Preferred Term 1 | Grade 1 | XX (XX.X) / XX |
| | Grade 2 | XX (XX.X) / XX |
| | Grade 3 | XX (XX.X) / XX |
| | Grade 4 | XX (XX.X) / XX |
| | Grade 5 | XX (XX.X) / XX |
| Preferred Term 2 | Grade 1 | XX (XX.X) / XX |
| | Grade 2 | XX (XX.X) / XX |
| | Grade 3 | XX (XX.X) / XX |
| | Grade 4 | XX (XX.X) / XX |
| | Grade 5 | XX (XX.X) / XX |
| | | ••• |
| System Organ Class 2 | Grade 1 | XX (XX.X) / XX |
| -1 5 | Grade 2 | XX (XX.X) / XX |
| | Grade 3 | XX (XX.X) / XX |
| | Grade 4 | XX (XX.X) / XX |
| | Grade 5 | XX (XX.X) / XX |



N: the number of patients in the Treated set (TS).

n: the number of patients with at least one TEAE within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

E: total number of TEAEs reported with appropriate severity.

For "Overall" and for each SOC and SOC/PT, each patient is counted once in the category of the maximum severity.

For "Overall", the number of all reported TEAEs are presented; for each SOC and SOC/PT, the number of TEAEs of maximum severity is given.

NCI CTCAE version 4.0 was used for assessing AE severity. AEs are coded using MedDRA version XX.X.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

< System organ classes (SOC) and preferred terms (PT) within each SOC should be sorted in descending order of n (%). >



Similar to table 3.7.1, the following tables will be constructed (with the corresponding corrections of underlined fragments in the note):

F. Hoffmann-La Roche Ltd MT.39355

Table 3.7.2 Treatment-emergent adverse events during rollover study by maximum severity

Treated set (TS, patients continuing in the rollover study)  $Page \ X \ of \ X$ 

F. Hoffmann-La Roche Ltd ML39355

Table 3.7.3 Treatment-emergent adverse events during whole study period by maximum severity

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.8.1 Treatment-emergent adverse events related to the study drug during treatment period by maximum severity

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.8.2 Treatment-emergent adverse events related to the study drug during rollover study by maximum severity

F. Hoffmann-La Roche Ltd

Table 3.8.3 Treatment-emergent adverse events related to the study drug during whole study period by maximum severity

Treated set (TS) Page X of X



Similar to table 3.3.1, the following tables will be constructed (with the corresponding corrections of underlined fragments in the note):

F. Hoffmann-La Roche Ltd ML39355

Table 3.9.1 Treatment-emergent adverse events of special interest during treatment period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

MT<sub>1</sub>39355

Table 3.9.2 Treatment-emergent adverse events of special interest during rollover study

Treated set (TS, patients continuing in the rollover study)  $Page \ X \ of \ X$ 

F. Hoffmann-La Roche Ltd

ML39355

Table 3.9.3 Treatment-emergent adverse events of special interest during whole study period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

MT<sub>1</sub>39355

Table 3.10.1 Treatment-emergent adverse events leading to death during treatment period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.10.2 Treatment-emergent adverse events leading to death during rollover study

Treated set (TS, patients continuing in the rollover study)

Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.10.3 Treatment-emergent adverse events leading to death during whole study period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

ML39355



Table 3.11.1 Treatment-emergent adverse events leading to discontinuation of study drug during treatment period

Treated set (TS)
Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.11.2 Treatment-emergent adverse events leading to discontinuation of study drug during rollover study

Treated set (TS, patients continuing in the rollover study)

Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.11.3 Treatment-emergent adverse events leading to discontinuation of study drug during whole study period

Treated set (TS)

Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.12.1 Treatment-emergent adverse events related to the study drug and leading to death during treatment period

Treated set (TS)

Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.12.2 Treatment-emergent adverse events related to the study drug and leading to death during rollover study

Treated set (TS, patients continuing in the rollover study)

Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.12.3 Treatment-emergent adverse events related to the study drug and leading to death during whole study period

Treated set (TS)

Page X of X

F. Hoffmann-La Roche Ltd

ML39355

Table 3.13.1 Non-serious treatment-emergent adverse events occurred at a frequency of >=5% during treatment period

Treated set (TS)

Page X of X

F. Hoffmann-La Roche Ltd



ML39355

Table 3.13.2 Non-serious treatment-emergent adverse events occurred at a frequency of >=5% during rollover study

Treated set (TS, patients continuing in the rollover study) Page X of X

F. Hoffmann-La Roche Ltd ML39355

Table 3.13.3 Non-serious treatment-emergent adverse events occurred at a frequency of >=5% during whole study period

Treated set (TS)
Page X of X



#### Table 3.14 Deaths

Treated set (TS)
Page X of X

| | Total |
|--------------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Total number of deaths | XX (XX.X) |
| Deaths during treatment period | XX (XX.X) |
| Deaths during rollover study | XX (XX.X) |

N: the number of patients in the Treated set (TS). n: the number of patients who died. Percentages are calculated as (100 x n/N).

Path to the program code, date and time of output



## **Pregnancies**

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.15 Urine pregnancy test

Treated set (TS)
Page X of X

| | Total |
|---------------------------------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Screening | |
| n' | XX |
| Done [1] | XX (XX.X) |
| Negative [2] | XX (XX.X) |
| Positive [2] | XX (XX.X) |
| Not Done [1] | XX (XX.X) |
| Male subject [1] | XX (XX.X) |
| Female subject with no childbearing potential [1] | XX (XX.X) |
| Other [1] | XX (XX.X) |
| Day 1 | |
| n' | XX |
| Done [1] | XX (XX.X) |
| Negative [2] | XX (XX.X) |
| Positive [2] | XX (XX.X) |
| Not Done [1] | XX (XX.X) |
| Male subject [1] | XX (XX.X) |
| Female subject with no childbearing potential [1] | XX (XX.X) |
| Other [1] | XX (XX.X) |
| ••• | ••• |

N: the number of women of childbearing potential in the TS. n' - the number of valid observations.

- n: the number of patients within a specific category.
- [1] Percentages are based on the corresponding number of valid observations.
- [2] Percentages are based on the number of patients for whom the pregnancy test was performed.

Path to the program code, date and time of output

<The following Urine pregnancy test assessments will be presented: Screening, Day 1, Week 4, Week 8, Week 12, Week 20, Week 26 Day 2>



## Laboratory tests

F. Hoffmann-La Roche Ltd ML39355

### Table 3.16 Hematology. Descriptive statistics

Treated set (TS)
Page X of X

Parameter: XXXXXXXXXXXXXXX, <units>

| | Total<br>(N = XX) | Change from the baseline |
|-----------|-------------------|--------------------------|
| Screening | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| MdX | AA | |
| Day 1 | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Max | ΔΛ | |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |

Data extracted: DD.MM.YYYY



### ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| ••• | | |
|-----|-------|-------|
| ••• | • • • | • • • |

N: the number of patients in the Treated set (TS).

n: the number of valid measurements.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug administration.

<The following assessments will be presented: Screening, Day 1, Baseline, Week 2, Week 4, Week 8, Week 16, Week 20, Week 26 Day 2, Follow-up visit, Week 39, Week 52>

<The following parameters will be presented: Leukocytes  $(10^9/L)$ , Erythrocytes  $(10^12/L)$ , Hemoglobin (g/L), Hematocrit (L/L), Platelets  $(10^9/L)$ ,
Neutrophils/Leukocytes (%), Eosinophils/Leukocytes (%), Basophils/Leukocytes (%), Monocytes/Leukocytes (%), Lymphocytes/Leukocytes (%).>

Path to the program code, date and time of output



Similar to table 3.16, the following tables will be constructed:

F. Hoffmann-La Roche Ltd
ML39355

Table 3.17 Blood chemistry. Descriptive statistics
Treated set (TS)
Page X of X

<The following parameters will be presented: Albumin (g/L), Alkaline Phosphatase (U/L), Alanine Aminotransferase (U/L), Aspartate Aminotransferase
(U/L), Direct bilirubin (umol/L), Bilirubin (umol/l), Protein (g/L), Cholesterol (mmol/L), Creatine Kinase (U/L), Creatinine (umol/L), Triglycerides
(mmol/L), Gamma Glutamyl Transferase (U/L), Glucose (mmol/L), Lactate Dehydrogenase (U/L), Calcium (mmol/L), Phosphate (mmol/L), Magnesium (mmol/L),
Potassium (mmol/L), Sodium (mmol/L), Urea nitrogen (mmol/L), Urate (umol/L), Creatinine Clearance (mL/min).>



F. Hoffmann-La Roche Ltd ML39355

#### Table 3.18 Hematology. Shift table

Treated set (TS)
Page X of X

Parameter: XXXXXXXXXXXXXXX, <units>

| | | Baseline | | |
|----------|-----------|-----------|-----------|-----------|
| | Low | Normal | High | Total |
| Baseline | | | | |
| Low | | | | XX (XX.X) |
| Normal | | | | XX (XX.X) |
| High | | | | XX (XX.X) |
| Total | | | | XX (100) |
| Week 2 | | | | |
| Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Week 4 | | | | |
| Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| ••• | | | | |
| • • • | ••• | • • • | • • • | • • • |

The baseline value for a variable is defined as the last non-missing value collected before the first study drug administration. Percentages are based on the number of patients with a non-missing assessment at the corresponding time point and at baseline.

<The following assessments will be presented: Baseline, Week 2, Week 4, Week 8, Week 16, Week 20, Week 26 Day 2, Follow-up visit, Week 39, Week 52>

Path to the program code, date and time of output



Similar to table 3.18, the following tables will be constructed:

F. Hoffmann-La Roche Ltd
ML39355

Table 3.19 Blood chemistry. Shift table
Treated set (TS)
Page X of X



F. Hoffmann-La Roche Ltd ML39355

### Table 3.20 Hematology. Out of range. Frequency table

Treated set (TS)
Page X of X

Parameter: XXXXXXXXXXXXX, <units>

| | Total |
|------------------|-------------------|
| | (N = XX)<br>n (%) |
| Screening | 1717 |
| n' | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| Day 1 | |
| n' | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| Baseline | |
| n' | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| Week 2 | |
| n' | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| • | |
| ••• | |
| ••• | ••• |

N: the number of patients in the Treated set (TS). n' - the number of valid observations.

<The following assessments will be presented: Screening, Day 1, Baseline, Week 2, Week 4, Week 8, Week 16, Week 20, Week 26 Day 2, Follow-up visit, Week 39, Week 52>

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.



Similar to table 3.20, the following tables will be constructed:

F. Hoffmann-La Roche Ltd
ML39355

Table 3.21 Blood chemistry. Out of range. Frequency table
Treated set (TS)
Page X of X



### Vital signs

F. Hoffmann-La Roche Ltd ML39355

### Table 3.22 Vital signs. Descriptive statistics

Treated set (TS)
Page X of X

Parameter: XXXXXXXXXXXXX, <units>

| | | Change from the baseline |
|-----------|-------|--------------------------|
| Screening | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Day 1 | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |

Data extracted: DD.MM.YYYY



### ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| •• | |
|-----|-------|
| ··· | • • • |

N: the number of patients in the Treated set (TS).

n: the number of valid measurements.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug administration.

Path to the program code, date and time of output

<Report all parameters: Systolic blood pressure, mm Hg/ Diastolic blood pressure, mm Hg/ Pulse rate, beats/minute/
Axillary temperature, C>

<The following assessments will be presented: Screening, Day 1, Baseline, Week 2, Week 4, Week 8, Week 16, Week 20, Week 26 Day 1, Week 26 Day 2, Follow-up visit, Week 39, Week 52>



F. Hoffmann-La Roche Ltd ML39355

### Table 3.23 Vital signs. Out of range. Frequency table

Treated set (TS)
Page X of X

Parameter: XXXXXXXXXXXXX, <units>

| | Total |
|------------------|-----------|
| | (N = XX) |
| | n (%) |
| Screening | |
| n' | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| Day 1 | |
| n' | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| Baseline | |
| n <b>'</b> | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| Week 2 | |
| n' | XX |
| Normal | XX (XX.X) |
| Out of Range NCS | XX (XX.X) |
| Out of Range CS | XX (XX.X) |
| ••• | |
| ••• | ••• |

N: the number of patients in the Treated set (TS). n' - the number of valid observations.

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.



Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

<Report all parameters: Systolic blood pressure, mm Hg/ Diastolic blood pressure, mm Hg/ Pulse rate, beats/minute/ Respiratory rate, breaths/minute/ Axillary temperature, C>

<The following assessments will be presented: Screening, Day 1, Baseline, Week 2, Week 4, Week 8, Week 16, Week 20, Week 26 Day 1, Week 26 Day 2, Follow-up visit, Week 39, Week 52>


# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

# Weight

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.24 Weight. Descriptive statistics

Treated set (TS)
Page X of X

Parameter: Weight, kg

| | Total $(N = XX)$ | Change from the baseline |
|-----------|------------------|--------------------------|
| Screening | | |
| n | XX | |
| Mean | XX.XX | |
| SD | XX.XXX | |
| Median | XX.XX | |
| Min | XX.X | |
| Max | XX.X | |
| Day 1 | | |
| n | XX | |
| Mean | XX.XX | |
| SD | XX.XXX | |
| Median | XX.XX | |
| Min | XX.X | |
| Max | XX.X | |
| Baseline | | |
| n | XX | |
| Mean | XX.XX | |
| SD | XX.XXX | |
| Median | XX.XX | |
| Min | XX.X | |
| Max | XX.X | |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX |
| Median | XX.XX | XX.XX |
| Min | XX.X | XX.X |
| Max | XX.X | XX.X |

Data extracted: DD.MM.YYYY



# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| ••• | | |
|-----|-------|-------|
| | • • • | • • • |

N: the number of patients in the Treated set (TS).

n: the number of valid measurements.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug administration.

Path to the program code, date and time of output

<The following assessments will be presented: Screening, Day 1, Baseline, Week 2, Week 4, Week 8, Week 16, Week 20, Week 26 Day 2, Follow-up visit>



# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

**ECG** 

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.25 ECG. Descriptive statistics

Treated set (TS)
Page X of X

Parameter: XXXXXXXXXXXXX, <units>

| | Total $(N = XX)$ | Change from the baseline |
|-----------|------------------|--------------------------|
| Screening | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Day 1 | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min | XX | |
| Max | XX | |
| Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |

Data extracted: DD.MM.YYYY



# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

| ••• | | |
|-------|-------|-------|
| • • • | ••• | • • • |
| | • • • | |

N: the number of patients in the Treated set (TS).

n: the number of valid measurements.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug administration.

Path to the program code, date and time of output

<Report all parameters: Heart rate, beats/min/ QT interval, ms/ QTC-F interval, ms>
<The following assessments will be presented: Screening, Day 1, Baseline, Week 4, Week 8, Week 26 Day 2, Week 52>



# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.26 ECG. Out of range and General assessment. Frequency table

Treated set (TS)
Page X of X

Parameter: XXXXXXXXXXXXXXXX

| | Total |
|--------------|-----------|
| | (N = XX) |
| | n (%) |
| Screening | |
| n' | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| Day 1 | |
| n' | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| Baseline | |
| n <b>'</b> | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| Week4 | |
| n' | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| <br> | |

N: the number of patients in the Treated set (TS). n' - the number of valid observations.

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.



Data extracted: DD.MM.YYYY



# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

Path to the program code, date and time of output

<Report all parameters: General assessment/ Heart rate, beats/min/ QT interval, ms/ QTC-F interval, ms>
<The following assessments will be presented: Screening, Day 1, Baseline, Week 4, Week 8, Week 26 Day 2, Week 52>



## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

# **Physical examinations**

F. Hoffmann-La Roche Ltd ML39355

#### Table 3.27 Physical examinations. Frequency table

Treated set (TS)
Page X of X

Body system: XXXXXXXXXXX

| | Total<br>(N = XX)<br>n (%) |
|--------------|----------------------------|
| Screening | |
| n' | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| Day 1 | |
| n' | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| Baseline | |
| n' | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| Week 2 | |
| n <b>'</b> | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |

N: the number of patients in the Treated set (TS).  $n^\prime$  - the number of valid observations.

n: the number of patients within a specific category. Percentages are based on the corresponding number of valid observations.



Data extracted: DD.MM.YYYY



Follow-up visit, Week 39, Week 52>

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

Path to the program code, date and time of output

<The following assessments will be presented: Screening, Day 1, Baseline, Week 2, Week 4, Week 8, Week 16, Week 20, Week 26 Day 1, Week 26 Day 2,</p>



## ML39355 STATISTICAL ANALYSIS PLAN Final 2.0 16 June 2020

## 16.2. Figures

No figures are planned in the study.

## 16.3. Listings

```
Listing 1 Disposition: analysis populations
Listing 2 Disposition: patient visits
Listing 3 Disposition: violation of inclusion/exclusion criteria
Listing 4 Disposition: study completion
Listing 5 Protocol deviations
Listing 6 Demographic and anthropometric characteristics
Listing 7 Baseline variables: Surgical lung biopsy (SLB)
Listing 8 Baseline variables: HRCT scan for patient eligibility confirmation
Listing 9 Baseline variables: Carbon monoxide diffusing capacity (DLCO)
Listing 10 Baseline variables: Pre- and post-bronchodilator spirometry parameters
Listing 11 Baseline variables: Serologic tests
Listing 12 Baseline variables: GAP assessment
Listing 13 Review transbronchial lung biopsy/Bronchoalveolar lavage (BAL)
Listing 14 General medical history
Listing 15 History of idiopathic pulmonary fibrosis (IPF)
Listing 16 Prior/concomitant medications
Listing 17 Prior/concomitant non-drug therapy and procedures
Listing 18 Spirometry
Listing 19 6-Minute Walk Test
Listing 20 Borg scale
Listing 21 EQ-5D questionnaire
Listing 22 HRCT scan
Listing 23 Adverse events
Listing 24 Exacerbations
Listing 25 Serious adverse events/Adverse events of special interest
Listing 26 Study drug administration
Listing 27 Exposure
Listing 28 Cases of incorrect administration of study drug / overdose
Listing 29 Urine pregnancy test
Listing 30 Hematology
Listing 31 Blood chemistry
Listing 32 Vital signs
Listing 33 ECG
Listing 34 Physical examinations
```

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 1 Disposition: analysis populations

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/<br>Race | Date, Time of informed consent signature | The Allocated to treatment set | Participation<br>in the<br>rollover<br>study | The<br>Treated<br>set (TS) | The Full<br>analysis<br>set (FAS) | Complete case<br>set (CCS) | Reason for<br>missing 26 week<br>FVC data | Treatment until Week 26 |
|---|---|---|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD<br>HH:MM | Yes | Yes | Yes | Yes | Yes | | Yes |
| XXXXXXXX/ X/<br>XX/ | YYYY-MM-DD<br>HH:MM | Yes | No | Yes | No | No | Death | No |
| XXXXXXX/ X/<br>XX/ | YYYY-MM-DD<br>HH:MM | No | No | No | No | No | Discontinuation<br>Lung<br>transplantation | No<br>No |

Path to the program code, date and time of output

Page 117 out of 151

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 2 Disposition: patient visits

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/<br>Race | Visit | Visit within visit window | Date / Study day | Main reason for unscheduled visit |
|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXXX | Yes | YYYY-MM-DD/ XX | |
| | XXXXXX | No | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | xxxxxxxxxx xxxxxxxxx |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 3 Disposition: violation of inclusion/exclusion criteria

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | Category | Criterion number/Criterion | Result |
|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | Inclusion criteria | xx/xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | No |
| | Exclusion criteria | XX/XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes |
| | Exclusion criteria | XX/XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes |
| | Eligibility confirmation | | No |
| • • • | | | |

Path to the program code, date and time of output

CONFIDENTIAL AND PROPRIETARY
Data MATRIX Ltd.

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 4 Disposition: study completion

All Enrolled patients
Page X of X

| Patient ID/ Sex/ Age<br>(years)/ Race | Date of study completion or discontinuation/ Study day | End of study status | Main reason for premature study termination |
|---|---|---|---|
| XXXXXXXX/ X/ XX/ XXXXX | YYYY-MM-DD/ XX | Discontinued | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXX/ X/ XX/ XXXXX | YYYY-MM-DD/ XX | Discontinued | Other: XXXXXXXXXXXXXXXXXXX |
| XXXXXXXX/ X/ XX/ XXXXX | YYYY-MM-DD/ XX | Completed | |
| XXXXXXX/ X/ XX/ XXXXX | YYYY-MM-DD/ XX | Screening failure | Presence or development of Inclusion/Exclusion criterion (-a): XXXXX |

. . .

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 5 Protocol deviations

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/ Race | Date of deviation<br>revealed / Study day | Visit name | Form name | Description of deviation |
|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD / XX | XXXXX | XXXXX | XXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD / XX | XXXXX | XXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD / XX | XXXXX | XXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| • • • | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 6 Demographics and anthropometric characteristics

All Patients Page X of X

| Patient ID/ | Date of birth | Age, years | Sex | Race | Ethnicity | Weight, kg | Height, cm | BMI, kg/m2 |
|---|---|---|---|---|---|---|---|---|
| Sex/ Age | | | | | | | | |
| (years)/ Race | | | | | | | | |
| XXXXXXX/ X/ | YYYY-MM-DD | XXXXX | XXXXX | XXXXX | XXXXX | XX | XXX | XX.X |
| XX/ XXXXX | | | | | | | | |
| XXXXXXX/ X/ | YYYY-MM-DD | XXXXX | XXXXX | XXXXX | XXXXX | XX | XXX | XX.X |
| XX/ XXXXX | | | | | | | | |
| XXXXXXX/ X/ | YYYY-MM-DD | XXXXX | XXXXX | XXXXX | XXXXX | XX | XXX | XX.X |
| XX/ XXXXX | | | | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 7 Baseline variables: Surgical lung biopsy (SLB)

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/ Race | Date of sample<br>collection/ Study<br>day | Assessment of regional specialist: UIP Pattern | Assessment of central specialist: UIP Pattern |
|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD/ XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD/ XX | XXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD/ XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ••• | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 8 Baseline variables: HRCT scan for patient eligibility confirmation

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | Date of HRCT scan/<br>Study day | Assessment of regional specialist: UIP Pattern | Assessment of central specialist (1): UIP Pattern | Assessment of central Reasons if Not Done specialist (2): UIP Pattern or Not performed |
|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/ XX | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxxx |
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/ XX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXX |
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/ XX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxxx |
| ••• | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 9 Baseline variables: Carbon monoxide diffusing capacity (DLCO)

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/ Race | Date, Time of<br>assessment/<br>Study day | Date, Time of<br>Hb assessment/<br>Study day | Hb value | Hb units | Parameter | DLCO result, % |
|---|---|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD HH:MM/ XX | | | | Predicted DLCO | XXXXX |
| | | YYYY-MM-DD<br>HH:MM/ XX | XX | XXXXX | Hb-corrected DLCO | XXXXX |
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD HH:MM/ XX | | | | Predicted DLCO | XXXXX |
| | | YYYY-MM-DD<br>HH:MM/ XX | XX | XXXXX | Hb-corrected DLCO | XXXXX |
| • • • | | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 10 Baseline variables: Pre- and post-bronchodilator spirometry parameters

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | Date of<br>assessment/<br>Study day | Time of assessment | Period of assessment | Parameter | Result | Units | Reason if Not Done |
|---|---|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/<br>XX | HH:MM | Before<br>bronchodilator<br>administration | FVC (absolute) | XXX | mL | |
| | | | | FVC (relative) predicted | XXX | % | |
| | | | | FEV1/FVC | XX.X | | |
| | | | : | ••• | • • • | _ | |
| | | HH:MM | After<br>bronchodilator<br>administration | FVC (absolute) | XXX | mL | |
| | | | | • • • | • • • | | |
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/<br>XX | нн:мм | Before<br>bronchodilator<br>administration | FVC (absolute) | Not Done | | XXXX XX XXXXXXXX |
| | | нн:мм | After<br>bronchodilator<br>administration | FVC (absolute) | XXX | mL | |
| | | | | • • • | • • • | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 11 Baseline variables: Serologic tests

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/ Race | Date, Time of<br>assessment/ Study<br>day | Lab Test | Fasting Status | Result | Reason if Not Done |
|---|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD HH:MM/<br>XX | Rheumatoid factor | Yes | XXXXX | |
| | | Anticyclic citrullinated peptide | Yes | XXXXX | |
| | | Antinuclear antibody titer | | Not Done | XXXXXXX XXXXXXXXXXX |
| XXXXXXXX/ X/ XX/<br>XXXXX | YYYY-MM-DD HH:MM/<br>XX | Rheumatoid factor | No | XXXXX | |
| | | Anticyclic citrullinated peptide | No | XXXXX | |
| | | Antinuclear antibody titer | No | XXXXX | |
| • • • | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 12 Baseline variables: GAP assessment

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/<br>Race | Date of<br>assessment/<br>Study day | FVC, %, predicted | Dlco, %,<br>predicted | Stage/<br>GAP Index | Mortality<br>(1-y) | Mortality<br>(2-y) | Mortality<br>(3-y) | Reason if Not<br>Done |
|---|---|---|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/ XX | XXXXX | XXXXX | X/XXXXX | XXXXX | XXXXX | XXXXX | XXXXXXXXX |
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/ XX | XXXXX | XXXXX | X/XXXXX | XXXXX | XXXXX | XXXXX | XXXXXXXXX |
| XXXXXXXX/ X/<br>XX/ XXXXX | YYYY-MM-DD/ XX | XXXXX | XXXXX | X/XXXXX | XXXXX | XXXXX | XXXXX | XXXXXXXXX |
| • • • | | | | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 13 Review transbronchial lung biopsy/ Bronchoalveolar lavage (BAL)

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/<br>Race | Visit | Medical procedure | Date of sample<br>collection/ Study<br>day | Are there features supporting an alternative diagnosis? | Comments if Yes | Result |
|---|---|---|---|---|---|---|
| XXXXXXXX/ X/ XX/ | XXXXXXX | Transbronchial biopsy | YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXX | | | | | XXXXXXX | |
| | | Bronchoalveolar | YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | lavage (BAL) | | | XXXXXX | |
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXXXX | Transbronchial biopsy | YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | Bronchoalveolar<br>lavage (BAL) | YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXXXX | Transbronchial biopsy | YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | Bronchoalveolar<br>lavage (BAL) | YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ••• | | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 14 General medical history

All Enrolled patients
Page X of X

| Patient ID/ | System Organ Class/ | Start Date / | End date / | Ongoing or | Comments |
|---|---|---|---|---|---|
| Sex/ Age | Preferred Term/ | Study day | Study day | Resolved | |
| (years)/ | Lowest Level Term/ | | | | |
| Race | Investigator Description | | | | |
| XXXXXXXX/ | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD/ XX | YYYY-MM-DD/ XX | Resolved | XXXXXXXXX |
| X/ XX/ | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |
| XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |

Terms are coded by MedDRA version XX.X.

Path to the program code, date and time of output

< Sort by start date, end date, SOC, PT, LLT>

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 15 History of idiopathic pulmonary fibrosis (IPF)

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | Diagnosis | Duration of clinical<br>symptoms consistent<br>with IPF (in months) | Clinically significant<br>environmental exposure<br>known to cause<br>pulmonary fibrosis | Known explanation for interstitial lung disease | Cigarette smoking<br>within 28 days before<br>the treatment start |
|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | Idiophatic Pulmonary Fibrosis | XX | Yes | No | Yes |
| XXXXXXXX/ X/<br>XX/ XXXXX | Idiophatic Pulmonary Fibrosis | XX | Yes | No | No |
| XXXXXXXX/ X/<br>XX/ XXXXX | Idiophatic Pulmonary Fibrosis | XX | No | Yes | Yes |
| ••• | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 16 Prior/concomitant medications

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/<br>Race | 1st Lvl, Anatomical main group/<br>2nd Lvl, Therapeutic subgroup/<br>3rd Lvl, Pharmacological subgroup/<br>4th Lvl, Chemical subgroup/<br>5th Lvl, Chemical substance/<br>Medication | Prior/<br>Concomitant | Start date, Time/<br>Study day/<br>Stop date, Time/<br>Study day | Dose (Units)/<br>Frequency/<br>Route | Indication for use | Comments |
|---|---|---|---|---|---|---|
| XXXXXXX/ X/<br>XX/ XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | P | YYYY-MM-DD HH:MM/ XX/<br>YYYY-MM-DD HH:MM/ XX | XXXXX (XXXXX) /<br>XXXXX/<br>XXXXX | XXXXXXXXXX | XXXXXXXXX |
| XXXXXXX/ X/<br>XX/ XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | С | YYYY-MM-DD HH:MM/ XX/<br>Ongoing | XXXXX (XXXXX) /<br>XXXXX/<br>XXXXX | XXXXXXXXXX | XXXXXXXXX |

P=Prior, C=Concomitant.

Medications are coded using WHODD version XX.X.

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 17 Prior/concomitant non-drug therapy and procedures

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/<br>Race | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/ | Prior/<br>Concomitant | Start date, Time/<br>Study day/<br>Stop date, Time/ | Indication | Comments |
|---|---|---|---|---|---|
| | Treatment | | Study day | | |
| XXXXXXXX/ X/ XX/ | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | P | YYYY-MM-DD HH:MM/ XX/ | XXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | YYYY-MM-DD HH:MM/ XX | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |

. . .

Non-drug therapy and procedures are coded using MedDRA version XX.X.

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

# Listing 18 Spirometry All Enrolled patients Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | Visit | Date, Time of<br>assessment/ Study<br>day | Parameter | Result | Units | Change from baseline/Base line | Reason if<br>Not Done |
|---|---|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | Screening/Retrospe ctive values | YYYY-MM-DD/ XX | FVC<br>(absolute) | XXXXX | mL | | |
| 7777 7777777 | ccive varues | | FVC | XXXXX | 용 | | |
| | | | (relative) | | Ü | | |
| | | | predicted | | | | |
| | | YYYY-MM-DD/ XX | FVC | XXXXX | mL | | |
| | | | (absolute) | | | | |
| | | | FVC | XXXXX | % | | |
| | | | (relative) | | | | |
| | | | predicted | | | | |
| | Screening | YYYY-MM-DD/ XX | FVC | XXXXX | mL | | |
| | screening | IIII-MM-DD/ XX | (absolute) | ΛΛΛΛΛ | Ш | | |
| | | | FVC | XXXXX | 용 | | |
| | | | (relative) | ΛΛΛΛΛ | 70 | | |
| | | | predicted | | | | |
| | Day 1 | YYYY-MM-DD HH:MM/ | FVC | XXXXX | mL | | |
| | Day 1 | XX | (absolute) | 71717171 | ш | | |
| | | 2121 | FVC | XXXXX | 용 | | |
| | | | (relative) | ********* | Ü | | |
| | | | predicted | | | | |
| | Week 12 | | FVC | Not | | | XXXXXXXXX |
| | | | (absolute) | Done | | | |
| | | YYYY-MM-DD HH:MM/ | FVC | XXXXX | % | XXXXX/XXXXX | |
| | | XX | (relative) | | | | |
| | | | predicted | | | | |
| | Week 26 | YYYY-MM-DD/ XX | FVC | XXXXX | mL | XXXXX/XXXXX | |
| | | | (absolute) | | | | |
| | | | FVC | XXXXX | 용 | XXXXX/XXXXX | |
| | | | (relative) | | | | |
| | | | predicted | | | | |
| | • • • | • • • | • • • | • • • | • • • | • • • | |
| • • • | | | | | | | |



# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

Path to the program code, date and time of output Data extracted: DD.MM.YYYY

<For screening list values before bronchodilator administration only.>

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 19 6-Minute Walk Test

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | Visit | Date of assessment /<br>Study day | Result, m | Change from<br>Baseline/Baseline | Reason if Not Done |
|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | XXXXX | YYYY-MM-DD / XX | XXXXX | XXXXX/XXXXX | |
| | XXXXX | YYYY-MM-DD / XX | XXXXX | XXXXX/XXXXX | |
| | XXXXX | YYYY-MM-DD / XX | XXXXX | XXXXX/XXXXX | |
| • • • | | | | | |

Path to the program code, date and time of output

Page 136 out of 151

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 20 Borg scale

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | Visit | Date of<br>assessment/<br>Study day | Timepoint | Time of assessment | Result | Change from Pre-<br>test Baseline/<br>Pre-test<br>Baseline | Change from<br>Baseline/<br>Baseline | Reason if Not<br>Done |
|---|---|---|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | XXXXX | YYYY-MM-DD/<br>XX | Before the 6-<br>minute exercise | HH:MM | XXXXX | | | |
| | | | After the 6-<br>minute exercise | HH:MM | XXXXX | XXXXX/XXXXX | | |
| | XXXXX<br>XX | YYYY-MM-DD/<br>XX | Before the 6-<br>minute exercise | HH:MM | XXXXX | | XXXXX/XXXXX | |
| | | | After the 6-<br>minute exercise | HH:MM | XXXXX | XXXXX/XXXXX | | |
| ••• | | | | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 21 EQ-5D-5L questionnaire

All Enrolled patients
Page X of X

| XXXXXXXXX | Patient ID/ Sex/<br>Age (years)/ Race | Visit | Date, Time of<br>assessment/<br>Study day | Mobility/ Self-care/ Usual activities/ Pain/Discomfort/ Anxiety/Depression | Your own health<br>state today<br>(VAS)/<br>Change from<br>Baseline/<br>Baseline | Index score/<br>Change from<br>Baseline/<br>Baseline | Reason if Not<br>Done |
|---|---|---|---|---|---|---|---|
| | | XXXXX | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX/XXXX/XXXX | XXXXX/XXXXX/XXXX | XXXXXXXXXXXXX |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

# Listing 22 HRCT scan All Enrolled patients

Page X of X

| Patient ID/ Sex/<br>Age (years)/ Race | Visit | Date of HRCT scan /<br>Study day | Parameter | Result | Change from<br>Baseline/Baseline | Reason if Not Done |
|---|---|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXX | YYYY-MM-DD / XX | HRCT fibrosis score | XXXXX | XXXXX/XXXXX | |
| | | | Ground-glass<br>opacity | XXXXX | XXXXX/XXXXX | |
| | XXXXX | YYYY-MM-DD / XX | HRCT fibrosis score | XXXXX | XXXXX/XXXXX | |
| | | | Ground-glass<br>opacity | Not Done | | XXXXXXXXXXXXXXXX |

Path to the program code, date and time of output

## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 23 Adverse events

All Enrolled patients Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/<br>Race | AE No/<br>TEAE<br>[1]/<br>SAE<br>[2] | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/<br>Reported Term | Start Date, Time/ Study Day/ End Date, Time/ Study Day/ Study period | Intermittent or persistent/ Severity/ Relationship to IMP/ Outcome | Action taken with IMP/ Concomitant medications?/ AESI?/ Exacerbation of IPF?/ Causality to concomitant medications taken |
|---|---|---|---|---|---|
| XXXXXXXX/ | XX/ | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/ XXX/ | XXXXXXXXXX/ | XXXXXXXXX/ |
| X/ XX/ | XXX/ | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/ XXX/ | XXXXXXXXX/ | XXX/ XXX/ XXX/ |
| XXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXX | XXXXXXXXX/ | XXXXXXXX, XXXXXXXXXXX, XXXXXXXXX |
| | (X, X) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | XXXXXXXXX | |

. . .

Abbreviations: AE = Adverse Event, SAE = Serious Adverse Event, TEAE = Treatment-Emergent Adverse Event.

Path to the program code, DDMMMYYYY, HH:MM

Date of data extraction: DDMMMYYYY

<sup>[1]</sup> TEAE is any reported adverse event that starts after initiation of the study therapy.

<sup>[2]</sup> Seriousness criteria: 1 = <<fatal>>, 2 = <<li>crequires or prolongs in-patient hospitalization>>, 4 = <<results in persistent or significant incapacity/disability>>, 5 = <<congenital abnormality or birth defect>>, 6 = <<other significant medical event>>.

AEs are coded using MedDRA version XX.X.

## ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 24 Exacerbations

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years)/ Race | AE No/<br>TEAE [1]/<br>SAE [2]/<br>Study<br>period | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/<br>Reported Term | Start Date, Time/<br>Study Day/<br>End Date, Time/<br>Study Day/ | Intermittent or persistent/<br>Severity/<br>Relationship to Study<br>Treatment/Outcome | Action taken with IMP/ Concomitant medications?/ AESI?/ Exacerbation of IPF?/ Causality to concomitant medications taken |
|---|---|---|---|---|---|
| XXXXXXXX/ X/<br>XX/ XXXXX | XX/<br>XXX/<br>XXX (X)/<br>XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/XXX/<br>YYYY-MM-DD HH:MM/XXX | XXXXXXXXX/XXXXXXXXX/<br>XXXXXXXXX/XXXXXXXX | XXXXXXXXX/<br>XXX/ XXX/ XXX/<br>XXXXXXXX, XXXXXXXXXX |

. . .

Abbreviations: AE = Adverse Event, SAE = Serious Adverse Event, TEAE = Treatment-Emergent Adverse Event.

Path to the program code, DDMMMYYYY, HH:MM

Date of data extraction: DDMMMYYYY

<sup>[1]</sup> TEAE is any reported adverse event that starts after initiation of the study therapy.

<sup>[2]</sup> Seriousness criteria: 1 = <<fatal>>, 2 = <<li>crequires or prolongs in-patient hospitalization>>, 4 = <<results in persistent or significant incapacity/disability>>, 5 = <<congenital abnormality or birth defect>>, 6 = <<other significant medical event>>.

Exacerbations are coded using MedDRA version XX.X.

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 25 Serious adverse events/Adverse events of special interest

All Enrolled patients
Page X of X

| Patient<br>ID/ Sex/<br>Age<br>(years)/<br>Race | SAE<br>No | Reported Term/<br>Date of Initial<br>SAE/AESI Report<br>Release/ Study Day | Report<br>type | Date event became<br>serious/ Study Day/<br>End date of<br>SAE/AESI/ Study Day/<br>Last dose prior to<br>SAE/AESI/ Study Day/ | Action taken due to<br>SAE/AESI/<br>Suspected causes | Description for Initial Report/<br>Description for Follow-up Report |
|---|---|---|---|---|---|---|
| XXXXXXXX/<br>X/ XX/<br>XXXXX | XX | XXXXXXXXXXX<br>XXXXXXXXXXXX<br>XXXXXXXXXX/<br>YYYY-MM-DD/XXX | Initial | YYYY-MM-DD/XXX/<br>YYYY-MM-DD/XXX/<br>YYYY-MM-DD/XXX | XXXXXXXXXX,<br>XXXXXXXXXX/<br>XXXXXXXXXX,<br>XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Abbreviations: SAE = Serious Adverse Event, AESI = AE of Special Interest. Terms are coded using MedDRA version XX.X.

Path to the program code, DDMMMYYYY, HH:MM

Date of data extraction: DDMMMYYYY

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

F. Hoffmann-La Roche Ltd ML39355

#### Listing 26 Study drug administration

Treated set (TS)
Page X of X

| Patient ID/ Sex/<br>Age (years)/ Race | Study period | Trade name | Single dose<br>(capsules)/<br>Frequency | Start Date/<br>Study day /<br>End Date / Study<br>day or Ongoing | Reason for dose<br>change or stop | Comments |
|---|---|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | Treatment period | Pirfenidone | XXXXX/<br>XXXXX | YYYY-MM-DD/ XX /<br>YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXX |
| | Treatment<br>period | Pirfenidone | XXXXX/<br>XXXXX | YYYY-MM-DD/ XX /<br>YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXX |
| | Rollover study | XXXXXXXXX | XXXXX/<br>XXXXX | YYYY-MM-DD/ XX /<br>YYYY-MM-DD/ XX | XXXXX | XXXXXXXXXXXXX |
| ••• | | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 27 Exposure

Treated set (TS)
Page X of X

| Patient ID/ Sex/ Age (years)/ Race | Study period | Duration of exposure, weeks | Number of capsules taken |
|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | Treatment period | XX.X | XXX |
| | Rollover study | XX.X | xxx |
| | Total | XX.X | xxx |
| ••• | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 28 Cases of incorrect administration of study drug / overdose

Treated set (TS)
Page X of X

| Patient ID/ Sex/ Age (years)/ Race | Study period | Date, Time/ Study day | Dose (capsules) | Category | Comments/Description |
|---|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXX | YYYY-MM-DD HH:MM/ XX | XXXXX | Incorrect administration of study drug | XXXXXXXXXXXXX |
| XXXXXXX/ X/ XX/<br>XXXXX | XXXXX | YYYY-MM-DD HH:MM/ XX | XXXXX | Incorrect<br>administration of<br>study drug | XXXXXXXXXXXXX |
| XXXXXXX/ X/ XX/<br>XXXXX<br> | XXXXX | YYYY-MM-DD HH:MM/ XX | XXXXX | Overdose | XXXXXXXXXXXXX |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 29 Urine pregnancy test

All Enrolled patients
Page X of X

| Patient ID/ Sex/<br>Age (years)/ Race | Visit | Date, Time of test<br>performed/ Study day | Result | Reasons if Not Done | _ |
|---|---|---|---|---|---|
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXX | YYYY-MM-DD HH:MM/ XX | XXXXX | | |
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXX | YYYY-MM-DD HH:MM/ XX | Not Done | xxxxxx xxxxxxxx xxxx | |
| XXXXXXXX/ X/ XX/<br>XXXXX | XXXXX | YYYY-MM-DD HH:MM/ XX | XXXXX | | |
| ••• | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 30 Hematology

All Enrolled patients
Page X of X

| Patient<br>ID/ Sex/<br>Age<br>(years) /<br>Race | Visit | Date,<br>Time of<br>specimen<br>collected<br>/ Study<br>day | Fasting<br>Status | Parameter,<br>units | Result | Units | Change from<br>Baseline/<br>Baseline | Reference<br>Limits<br>Lower/Upper | Out of<br>Range<br>(L/N/H) | CS (Yes/No) | Reason<br>if Not<br>Done |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXX/<br>X/ XX/<br>XXXXX | XXXXX | YYYY-MM-<br>DD HH:MM/<br>XX | Yes | XXXXX | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX/XXXXX | X | XXXXX | |
| | | | | XXXXX | Not Done | | | | | | XXXXXXX |
| | | | | XXXXX | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX/XXXXX | X | XXXXX | |
| | XXXXX | YYYY-MM-<br>DD HH:MM/<br>XX | Yes | XXXXX | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX/XXXXX | X | XXXXX | |
| | ••• | | | | | | | | | | |

L = below lower reference limit. H = above upper reference limit. N = Normal range. CS = Clinically Significant.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 31 Blood chemistry

All Enrolled patients
Page X of X

| Patient<br>ID/ Sex/<br>Age<br>(years) /<br>Race | Visit | Date, Time of specimen collected / Study day | Fasting<br>Status | Parameter,<br>units | Result | Units | Change from<br>Baseline/<br>Baseline | Reference<br>Limits<br>Lower/Upper | Out of<br>Range<br>(L/N/H) | CS (Yes/No) | Reason<br>if Not<br>Done |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXX/<br>X/ XX/<br>XXXXX | XXXXX | YYYY-MM-<br>DD HH:MM/<br>XX | Yes | XXXXX | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX/XXXXX | X | XXXXX | |
| | | | | XXXXX | Not Done | | | | | | XXXXXXXX<br>XXXXX |
| | | | | XXXXX | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX/XXXXX | X | XXXXX | |
| | XXXXX | YYYY-MM-<br>DD HH:MM/<br>XX | Yes | XXXXX | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX/XXXXX | X | XXXXX | |
| | • • • | | | | | | | | | | |

L = below lower reference limit. H = above upper reference limit. N = Normal range. CS = Clinically Significant.

Path to the program code, date and time of output

Data extracted: DD.MM.YYYY

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

# Listing 32 Vital signs All Enrolled patients

Page X of X

| Patient ID/<br>Sex/ Age<br>(years) / | Visit | Date, Time of assessment/ | Parameter | Result | Units | Change from<br>Baseline/<br>Baseline | Out of<br>Range<br>(Yes/No) | Clinically<br>Significant<br>(Yes/No) | Reason if Not<br>Done |
|---|---|---|---|---|---|---|---|---|---|
| Race | | Study day | | | | | | | |
| XXXXXXXXX/<br>X/ XX/ XXXXX | XXXXX | YYYY-MM-DD<br>HH:MM/ XX | Systolic Blood<br>Pressure | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Diastolic Blood<br>Pressure | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Pulse rate | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Respiratory rate | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Axillary<br>temperature | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Weight | XXXXX | XXXXX | XXXXX/XXXXX | | | |
| | | | BMI | XXXXX | XXXXX | XXXXX/XXXXX | | | |
| | | | Height | XXXXX | XXXXX | | | | |
| | XXXXX | YYYY-MM-DD<br>HH:MM/ XX | Systolic Blood<br>Pressure | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Diastolic Blood<br>Pressure | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Pulse rate | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Respiratory rate | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Axillary<br>temperature | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | Weight<br>BMI | XXXXX | XXXXX | XXXXX/XXXXX | | | |
| | | | Height | XXXXX | XXXXX | | | | XXXXXXXXXXXXX |
| | | • • • | | | | | | | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 33 ECG

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years) /<br>Race | Visit | Date, Time<br>of<br>assessment /<br>Study day | Parameter | Result | Units | Change from<br>Baseline/<br>Baseline | Out of<br>Range<br>(Yes/No) | Clinically<br>Significant<br>(Yes/No) | Reason /<br>Comments if<br>Not Done /<br>Abnormal |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXXX/ X/<br>XX/ XXXXX | XXXXX | YYYY-MM-DD<br>HH:MM/ XX | Heart rate | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | QT interval | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | QTC-F interval | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | General assessment | XXXXX | | | | XXXXX | |
| | XXXXX | YYYY-MM-DD | Heart rate | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | HH:MM/ XX | QT interval | Not Done | | | | | XXXXXXX XXXX |
| | | | QTC-F interval | XXXXX | XXXXX | XXXXX/XXXXX | XXXXX | XXXXX | |
| | | | General assessment | XXXXX | | | | XXXXX | |

Path to the program code, date and time of output

# ML39355\_STATISTICAL ANALYSIS PLAN\_Final 2.0\_17 June 2020

F. Hoffmann-La Roche Ltd ML39355

#### Listing 34 Physical examinations

All Enrolled patients
Page X of X

| Patient ID/<br>Sex/ Age<br>(years) / Race | Visit | Date, Time<br>of<br>assessment /<br>Study day | Body system/Site | Result | Clinically<br>Significant<br>(Yes/No) | Reason/ Comments if Not Done/<br>Abnormal |
|---|---|---|---|---|---|---|
| XXXXXXXXX/ X/<br>XX/ XXXXX | XXXXX | YYYY-MM-DD<br>HH:MM/ XX | Head | XXXXX | XXXXX | |
| | | | Eyes | XXXXX | XXXXX | |
| | | | Ears, nose and throat | XXXXX | XXXXX | |
| | | | Cardiovascular system | Not Done | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | Dermatological system | XXXXX | XXXXX | |
| | | | Musculoskeletal system | XXXXX | XXXXX | |
| | | | • • • | XXXXX | XXXXX | |
| XXXXXXXXX/ X/<br>XX/ XXXXX | XXXXX | YYYY-MM-DD<br>HH:MM/ XX | Head | XXXXX | XXXXX | |
| | | | Eyes | XXXXX | XXXXX | |
| | | | Ears, nose and throat | XXXXX | XXXXX | |
| | | | Cardiovascular system | XXXXX | XXXXX | |
| | | | Dermatological system | XXXXX | XXXXX | |
| | | | Musculoskeletal system | XXXXX | XXXXX | |
| | | | • • • | XXXXX | XXXXX | |
| ••• | | | | | | |

Path to the program code, date and time of output